Protocol: BCX4430-106-DMID18-0013

Version Date: 10-April-2019

# Statistical Analysis Plan

Sponsor: BioCryst Pharmaceuticals, Inc.

Protocol No: BCX4430-106-DMID18-0013

Protocol Title: A phase 1 double-blind, placebo-controlled, dose-ranging study to evaluate the safety, tolerability, and pharmacokinetics of galidesivir (BCX4430) administered as single doses via intravenous infusion in healthy subjects

PRA Project ID: BIO139GF-181392


# **Approvals**

The undersigned have approved this Statistical Analysis Plan for use in this study.

| Name of Sponsor<br>Representative / Title: | Sharon C. Murray, PhD / Director Biostatistics, BioCryst Pharmaceuticals |
|---|---|
| Signature of Sponsor<br>Representative / Date: | Shown C. Wherrow 16APR 2019 |
| Name of Sponsor<br>Representative / Title: | Diane Gesty-Palmer, MD / Senior Medical Director, BioCryst Pharmaceuticals |
| Signature of Sponsor Representative / Date: | Diamen Polne 16 APR 2019. |
| Name of Sponsor<br>Representative / Title | Elliott Berger, MD / Senior Vice President, Regulatory Affairs, BioCryst Pharmaceuticals |
| Signature of Sponsor<br>Representative / Date: | Devilley 16 APRIL 2015 |
| Name of Sponsor<br>Representative / Title: | Amanda Mathis, PhD / Director of Clinical Pharmacology |
| Signature of Sponsor<br>Representative / Date: | amanda Mallon 16april 2019 |
| Name of Author / Title: | Jacqueline Cater / Senior Biostatistician, PRA Health Sciences |
| Signature of Author / Date: | Cornellay Chap to gain to a complete the complete that the complet |



# **Table of Contents**

| Approvals | |
|-------------------------------------------------------|----|
| Table of Contents | |
| 3.0 Introduction | 4 |
| 4.0 Changes from Previous Version of Approved SAP | |
| 5.0 Study Objectives | |
| 5.1 Primary Objective | 4 |
| 5.1.1 Primary Endpoints | 4 |
| 5.2 Secondary Objective | 4 |
| 5.2.1 Secondary Endpoints | 4 |
| 6.0 Study Design | |
| 6.1 Sample Size Considerations | 6 |
| 6.2 Randomization | |
| 7.0 Overview of Planned Analysis | |
| 7.1 Changes from Protocol | |
| 7.2 Interim Analysis and Key Results | |
| 7.3 Final Analysis | |
| 8.0 Data Review | |
| 8.1 Data Management | |
| 8.2 Acceptance of Data for Summarization | |
| 9.0 Definitions and General Analysis Methods | |
| 9.1 Analysis Data Presentation | |
| 9.1.1 Rounding | |
| 9.1.2 Imputation | |
| 9.1.3 Descriptive Statistics | |
| 9.1.4 Pooling | |
| 9.1.5 Unscheduled Measurements | و |
| 9.2 Analysis Data Definitions | |
| 9.2.1 Baseline Definition | |
| 9.2.2 Treatment/Subject Grouping | |
| 9.2.3 Common Variable Derivations | |
| 9.2.4 QC | |
| 9.2.5 ADaM Datasets and Metadata | |
| 9.3 Software | |
| 9.4 Statistical Methods | |
| 9.4.1 Statistical Outlier Determination | |
| 9.4.2 Predetermined Covariates and Prognostic Factors | |
| 9.4.3 Hypothesis Testing | |
| 9.4.3.1 Primary Objective | |
| 9.4.3.2 Secondary Objective - Dose Proportionality | 10 |
| 9.5 TFL Layout | |
| 10.0 Analysis Populations | |
| 10.1 Safety Population | |
| 10.2 Pharmacokinetic Population | |
| 11.0 Subject Disposition | |
| 12.0 Protocol Deviations | |
| 13.0 Demographic and Baseline Characteristics | |
| 13.1 Demographics | |
| 13.2 Medical History | |
| 13.3 Screening Results | |
| 14.0 Prior and Concomitant Medications | |
| 15.0 Treatment Exposure | |
| 16.0 Pharmacokinetic Variables | 13 |
| 16.1.1 Plasma Variables | |


| 16.1.2 Urine Variables | 14 |
|-----------------------------------------------------------------------|----|
| 16.2 Pharmacokinetic Summaries | 15 |
| 16.2.1 Plasma Concentrations | 15 |
| 16.2.2 Plasma Pharmacokinetic Parameters | 15 |
| 16.2.3 Urine Pharmacokinetic Parameters | 16 |
| 16.2.4 Dose Proportionality Analyses | 16 |
| 17.0 Safety Analyses | |
| 17.1 Safety Variables | |
| 17.1.1 Adverse Events | |
| 17.1.2 Deaths and Serious Adverse Events | 18 |
| 17.1.3 Laboratory Data | 18 |
| 17.1.4 Vital Signs | 19 |
| 17.1.5 Electrocardiograms | 19 |
| 17.1.6 Cardiac Telemetry | 19 |
| 17.1.7 Echocardiograms | |
| 17.1.8 Physical Examination | 19 |
| References | 20 |
| Appendix 1: Glossary of Abbreviations | 21 |
| Appendix 2: Schedules of Assessments from Protocol | 23 |
| Appendix 3: List of End of Text Outputs | |
| Appendix 4: Shells for Post-Text Tables, Figures and Listings | 29 |
| Appendix 5: Toxicity Table - Modified DMID Adult toxicity Table, 2014 | 29 |
| Document History | 35 |

Protocol: BCX4430-106-DMID18-0013


# 3.0 Introduction

This Statistical Analysis Plan (SAP) describes the statistical methods that will be used during the analysis and reporting of data collected under BioCryst Pharmaceuticals, Inc., Protocol BCX4430-106.

This SAP should be read in conjunction with the study protocol and electronic case report form (eCRF). This version of the SAP has been developed using the protocol dated 11-Jan-2019 and the final eCRF(s) dated 30-Oct-2018.

An approved and signed SAP is a requirement for database lock.

This SAP covers all results that will be processed by the PRA Early Development Services (EDS) Biostatistics Department.

PRA EDS will perform the final pharmacokinetic (PK) and safety and tolerability analyses.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they are identified. Any post-hoc or unplanned analyses, or substantive changes from the planned analysis in this SAP performed to provide results for inclusion in the clinical study report (CSR), will be clearly identified in the CSR. Changes to planned analyses do not require an updated SAP but should be denoted in the CSR if significant.

# 4.0 Changes from Previous Version of Approved SAP

Not applicable. This is the first version of the SAP.

# 5.0 Study Objectives

# 5.1 Primary Objective

The primary objective of the study is:

To evaluate the safety and tolerability of single ascending doses (SAD) of galidesivir (BCX4430) administered by intravenous (IV) infusion in healthy subjects.

## 5.1.1 Primary Endpoints

The primary endpoints of the study are:

 Safety and tolerability parameters including adverse events (AEs) and serious adverse events (SAEs), laboratory abnormalities, vital signs, electrocardiograms (ECGs), echocardiograms (ECHOs), cardiac telemetry, and physical examination (PE).

# 5.2 Secondary Objective

The secondary objective of the study is:

 To characterize the plasma pharmacokinetic (PK) profile and urinary elimination of SAD of galidesivir administered by IV infusion in healthy subjects.

# 5.2.1 Secondary Endpoints

The secondary endpoints of this study are:

The PK parameters for galidesivir, including: maximum concentration (C<sub>max</sub>), last measurable concentration of drug (C<sub>last</sub>), time to maximum concentration (T<sub>max</sub>), area under the concentration time curve from time zero to last time (AUC<sub>last</sub>), area under the concentration time curve from time zero to infinity (AUC<sub>inf</sub>), clearance (CL), volume of distribution (V<sub>z</sub>), percentage of AUC extrapolated between AUC<sub>last</sub> and AUC<sub>inf</sub> (AUC<sub>extrap</sub>), λ<sub>z</sub>, and half-life (t<sub>1/2</sub>), and other parameters, where appropriate.

EDSREP 009 T 01 G 


Dose proportionality of galidesivir based upon AUC<sub>inf</sub>, AUC from time 0 to time "t" (AUC<sub>t</sub>), and C<sub>max</sub>.

#### 6.0 Study Design

This SAD study will evaluate the safety, tolerability, and PK of single doses of galidesivir vs. placebo administered as IV infusions in healthy subjects enrolled in up to four dose cohorts of 8 subjects each, for a total of 32 subjects. A single dose of study drug will be administered per cohort: 6 subjects will receive galidesivir IV, and 2 subjects will receive matching placebo.

The planned cohorts are as follows:

- Cohort 1, Regimen A: 5 mg/kg galidesivir or placebo, IV infusion × 1 dose
- Cohort 2, Regimen B: 10 mg/kg galidesivir or placebo, IV infusion × 1 dose
- Cohort 3, Regimen C: 15 mg/kg galidesivir or placebo, IV infusion × 1 dose
- Cohort 4, Regimen D: 20 mg/kg galidesivir or placebo, IV infusion × 1 dose

Subjects will be randomized within each cohort to receive either galidesivir or placebo. As a safety precaution, on the first day of dosing in each cohort, only 2 subjects will be dosed (to be referred to as sentinel subjects). The randomization schedule will be constructed such that 1 of the sentinel subjects dosed on the first day will be randomized to receive galidesivir and 1 will be randomized to receive placebo. After review of the safety data from the 24-hour post-dose period for the sentinel subjects, which includes review of any AEs, any abnormalities in the bedside ECGs, safety laboratory assessments and vital signs, the remainder of the cohort (5 subjects randomized to galidesivir; 1 randomized to placebo) will be dosed at least 2 days after the sentinel subjects.

Enrollment of subjects in each sequential higher dose level cohort will occur only after completion of a clinical safety review of laboratory, AE, vital sign, ECG (12-lead and telemetry), and PE data for all subjects up through 96 hours post-dose and plasma PK data through 24 hours post-dose. Based upon safety review and evaluation of the data for each subject, adjustments in the dose escalation scheme for the next cohort may be made, including omission of higher dose cohorts in the event that the safety and PK parameters have been adequately characterized with lower dose cohorts. Where considered appropriate to meet the study objectives, adjustments in the protocol-specified dose escalation for subsequent cohorts are permissible (i.e., an intermediate dose between the previous tolerable dose and the scheduled next higher dose). The study design is shown in Figure 1 (below).

EDSREP 009 T 01 G 



Protocol: BCX4430-106-DMID18-0013 Version Date: 10-April-2019

Figure 1 BCX4430-106 Study Design



Abbreviations: D = day; PK = pharmacokinetic.

# 6.1 Sample Size Considerations

No formal power or sample size calculations were used to determine cohort sizes. Cohort sizes were based upon experience in other SAD Phase 1 studies. A sample size of 6 subjects receiving active drug per cohort should provide adequate characterization of PK and safety assessments within this setting.

#### 6.2 Randomization

This is a double-blind study; treatment assignment within a cohort will be blinded to the PI, clinical staff, study subjects, and the data management team, with the exception of the unblinded dosing team, if required. The randomization schedules will be generated by an unblinded study statistician. A computergenerated randomization schedule will be used to randomly assign subjects to galidesivir or placebo. Subjects in each of the Cohorts 1 to 4 will be randomized to galidesivir or placebo in a 3:1 ratio (ie, 6 subjects per cohort will be randomly assigned to receive galidesivir and 2 subjects per cohort will be randomly assigned to receive placebo). As a safety precaution, on the first day of dosing in all cohorts, 2 sentinel subjects will be initially dosed, and the randomization schedule will be generated so that in each cohort 1 sentinel subject is randomly assigned to receive galidesivir and 1 sentinel subject is randomly assigned to receive placebo. The remainder of the cohort will be randomized such that 5 subjects are assigned to receive galidesivir and 1 subject assigned to receive placebo.



Protocol: BCX4430-106-DMID18-0013 Version Date: 10-April-2019

Following confirmation of eligibility, subjects will be identified by a unique 5-digit subject identifier (e.g., 11001) in which the first digit indicates the study site identifier, the second digit indicates the cohort number and the final 3 digits indicate the subject number. Any replacement subjects will be identified by replacing the third digit "0" with "9". For example, if Subject 11005 withdraws from the study early, the replacement subject will be numbered 11905 and will receive the same study treatment (i.e., active or placebo) as Subject 11005.

Subject numbers will be as follows:

| Cohort | Subject Numbers | Replacement Subject Numbers |
|--------|-----------------|-----------------------------|
| 1 | 11001 to 11008 | 11901 to 11908 |
| 2 | 12001 to 12008 | 12901 to 12908 |
| 3 | 13001 to 13008 | 13901 to 13908 |
| 4 | 14001 to 14008 | 14901 to 14908 |

# 7.0 Overview of Planned Analysis

# 7.1 Changes from Protocol

There are no changes from the protocol.

# 7.2 Interim Analysis and Key Results

An interim PK report will be prepared by Biocryst for review by the DEC that will document the following PK findings for each dose cohort:

- Preliminary plasma PK parameters (through 24-hours post-dose) based upon nominal times: AUC; C<sub>max</sub>, T<sub>max</sub>, terminal elimination half-life (t<sub>1/2</sub>; median, minimum, maximum, geometric mean, coefficient of variation [CV%])
- Predictions of C<sub>max</sub> and AUC values for the next cohort, where relevant

# 7.3 Final Analysis

Draft TFLs will be provided after database lock. After Sponsor comments have been incorporated, the TFLs will be finalized and incorporated into the first draft of the CSR.

# 8.0 Data Review

# 8.1 Data Management

Data handling and transfer will take place under the PRA Data Management Plan for the study.

# 8.2 Acceptance of Data for Summarization

Programming of analysis datasets and TFLs may be ongoing during the data management of the study. However, programming of analysis datasets and TFLs will be completed and quality controlled (QC'd) after

EDSREP 009 T 01 G 


database lock. Only quality-assured results released by the Safety Laboratory, Bioanalytical Laboratory, or other external data source will be used for the programming of analysis datasets and TFLs for the final report. Any data values requiring investigation or corrections that are identified while programming the analysis datasets and TFLs will be sent to the project Data Manager. If the issue affects the TFLs the Programmer or Statistician who identified the issue will follow it to resolution.

# 9.0 Definitions and General Analysis Methods

# 9.1 Analysis Data Presentation

# 9.1.1 Rounding

In listings, data will be presented with the same precision as the original data. Derived data will be rounded for presentation purposes.

For all summaries, minimum (min) and maximum (max) will be presented to the same number of decimal places as the original data, the mean and median to 1 decimal greater than the original data, and the standard deviation (SD) to 2 decimals greater than the original data. Frequency percentages and percent coefficient of variation (CV%) will be presented to 1 decimal.

PK parameters will be rounded in the derived datasets as determined by the pharmacokineticist and presented as such in the listings. Each parameter will have a fixed number of decimals ( $C_{max}$  and AUC will have 3 significant figures, and half-life and  $T_{max}$  will have 1 decimal). In general, the pharmacokineticist will use discretion when deciding the number of decimals for each parameter.

### 9.1.2 Imputation

Unless otherwise noted, data will not be imputed.

#### 9.1.3 Descriptive Statistics

Unless otherwise indicated, continuous variables will be summarized with the following descriptive statistics: n (number of observations), (arithmetic) mean, SD, min, median, and max.

Categorical data will be summarized with frequencies and percentages. Percentages by categories will be based on the number of subjects exposed within a treatment. Percentages will be rounded to 1 decimal, except 100% which will be displayed without any decimal places. Percentages will not be displayed for zero counts. Categories will be presented in the tables exactly as they appear in the eCRF / database.

#### 9.1.4 Pooling

Placebo subjects will be pooled for summary TFLs for this study.

#### 9.1.5 Unscheduled Measurements

Unscheduled measurements will be included in the listings. In general, except for unscheduled measurements used for baseline, unscheduled measurements will be excluded from the descriptive statistics and statistical analysis by timepoint. For shift tables or tables that summarize worst outcome, unscheduled measurements (occurring after previous timepoint and up to and including each scheduled timepoint) will be included in summary statistics.

# 9.2 Analysis Data Definitions

#### 9.2.1 Baseline Definition

Unless otherwise stated, baseline for post dose evaluations is defined as the last observation recorded before the first study drug administration for each regimen as indicated in Appendix 2 (Schedule of Assessments). The last observation can be an unscheduled/repeated measurement. Baseline ECGs will

EDSREP 009 T 01 G 





be calculated from an average of the triplicate readings prior to initiation of treatment on Day 1 of each treatment period.

# 9.2.2 Treatment/Subject Grouping

Throughout this SAP, study drug refers to: BCX4430 galidesivir for IV infusion.

| Label | Grouping |
|---|---|
| Study Drugs | BCX4430 galidesivir for IV infusion |
| Treatment | Cohort 1: Regimen A: Galidesivir (Dose 5 mg/kg, Calculated Dose Range 250-500 mg, Concentration 1.0 mg/mL, Dose Volume 250-500 mL), or Placebo (Dose Volume 250-500 mL) |
| | <ul> <li>Cohort 2:</li> <li>Regimen B: Galidesivir (Dose 10 mg/kg, Calculated Dose Range 500-1000 mg, Concentration 1.0-2.0 mg/mL, Dose Volume 500 mL), or</li> <li>Placebo (Dose Volume 500 mL)</li> </ul> |
| | <ul> <li>Cohort 3:</li> <li>Regimen C: Galidesivir (Dose 15 mg/kg, Calculated Dose Range 750-1500 mg, Concentration 1.5-3.0 mg/mL, Dose Volume 500 mL), or</li> <li>Placebo (Dose Volume 500 mL)</li> </ul> |
| | Cohort 4: Regimen D: Galidesivir (Dose 20 mg/kg, Calculated Dose Range 1000-2000 mg, Concentration 2.0-4.0 mg/mL, Dose Volume 500 mL), or Placebo (Dose Volume 500 mL) |
| Dose Levels | BCX4430: 5 mg/kg, Calculated Dose Range 250-500 mg BCX4430: 10 mg/kg, Calculated Dose Range 500-1000 mg BCX4430: 15 mg/kg, Calculated Dose Range 750-1500 mg BCX4430: 20 mg/kg, Calculated Dose Range 1000-2000 mg [Note: Treatment labels will use mg/kg] |

# 9.2.3 Common Variable Derivations

| Variable | Data Type | Definition/Calculation |
|---|---|---|
| Change from baseline | All | Post-dose observation minus baseline observation |
| Analysis study day (prior to dose) | All | Date of measurement minus dose date |
| Analysis study day (post dose) | All | Date of measurement minus dose date + 1 |
| TEAE | AE | An AE is a treatment-emergent adverse event (TEAE) if the AE start date/time is greater than or equal to the first dose date/time |

Abbreviations: AE = adverse event; TEAE = treatment-emergent adverse event.

 EDSREP 009 T 01 G


#### 9.2.4 QC

The analysis datasets and the TFLs will be QC'd according to the PRA EDS QC plan.

#### 9.2.4.1 Critical Data

The QC plan requires datasets be classified as critical or non-critical. As the primary and secondary objectives of this study are to characterize the safety and tolerability of galidesivir as well as PK profile, critical datasets include subject level demographics, PK parameters, concentrations, and AEs.

#### 9.2.5 ADaM Datasets and Metadata

The analysis datasets will be generated in accordance with Clinical Data Interchange Standard Consortium (CDISC) Analysis Data Model (ADaM) Version 2.1.

ADaM-compliant datasets will be delivered to the sponsor. A define.xml file Version 2 with the corresponding metadata will be included. Analysis results metadata are excluded.

#### 9.3 Software

The statistical analysis and reporting will be done using SAS® for Windows™ Version 9.4 or higher (SAS Institute, Inc.).

PK parameter calculations will primarily be done using Phoenix® WinNonlin® Version 8.1 or higher (Certara, Inc.). Additional PK computations may be performed in SAS.

#### 9.4 Statistical Methods

#### 9.4.1 Statistical Outlier Determination

No statistical outlier analysis is planned.

#### 9.4.2 Predetermined Covariates and Prognostic Factors

There are no predetermined covariates or prognostic factors.

#### 9.4.3 Hypothesis Testing

#### 9.4.3.1 Primary Objective

No formal study hypothesis will be stated or tested in this Phase I study.

# 9.4.3.2 Secondary Objective - Dose Proportionality

Dose proportionality for  $AUC_{inf}$ ,  $AUC_{t}$ , and  $C_{max}$  will be evaluated using the power model (including all doses) and also using an ANOVA model where each dose will be compared with a reference dose in a pairwise basis. The mean slope from the power model and the set of pairwise comparisons from the ANOVA method will constitute descriptive evaluations of dose proportionality.

#### **Power Model**

The power model is as follows:

#### Equation 1:

$$log(Y_{ik}) = S_i^{[1]} + \beta \times log(Dose_k) + \epsilon_{ik}$$

where  $Y_{ik}$  is the measured response variable, AUC<sub>inf</sub>, AUC<sub>t</sub>, and  $C_{max}$ , on the  $k^{th}$  dose,  $S_{\ell}^{11}$  is random subject effect for the  $i^{th}$  subject, and  $\epsilon_{ik}$  is the random error. After exponentiation, the model equation 1 is identical to equation 2 (below).

EDSREP 009 T 01 G 





# Equation 2:

 $Y_{ik} = \alpha \times Dose^{\beta}$ 

where a includes the error.

Dose proportionality for PK parameters will be assessed by restricted maximum likelihood using SAS PROC MIXED. The mean slope will be estimated from the power model and the corresponding 90% CI calculated. If the 90% CI of the slope of the C<sub>max</sub> and AUCs contains 1, then dose proportionality is indicated.

#### Analysis of Variance

Following log-e transformation, dose-normalized PK parameters will be analyzed with an ANOVA model using PROC MIXED. Each dose will be compared with a reference dose on a pairwise basis. The ratio of geometric least squares means (LSM) and the corresponding 90% CI will be estimated for each PK parameter of interest. If the 90% CI for the geometric LSM ratio for a given pairwise comparison falls completely within the 0.8 to 1.25 equivalence region then dose proportionality is indicated.

# 9.5 TFL Layout

Report layout will be according to the PRA EDS standards, which are International Council for Harmonisation (ICH) E3 compliant. The layout of TFLs will be according to the PRA EDS standards.

TFL shells are provided with and approved as part of this SAP. Small changes to shell layout due to the nature of the data may be required after database lock at the discretion of the PRA project statistician. Other changes to the shells may be out of scope. The TFLs will be provided both individually in revisable text format (RTF) format, with separate files for each table, figure, and listing, and combined in Adobe PDF format. All TFLs will be in letter format.

# 10.0 Analysis Populations

| Analyses | Safety Population | PK Population |
|-------------------------------|-------------------|---------------|
| Disposition Summaries | ✓ | |
| Baseline Characteristics | <i>✓</i> | ✓ |
| Safety Assessments | <b>✓</b> | |
| Plasma Concentrations | · | |
| Plasma PK Parameters | | <b>✓</b> |
| Urine PK Parameters | | ✓ |
| Dose proportionality Analyses | | <b>√</b> |

# 10.1 Safety Population

The safety population will include all randomized subjects who received any amount of study drug (ie, a partial infusion). Subjects will be analyzed according to the treatment received. This population will be used for all analyses of accountability, demographics, galidesivir drug concentration, and safety.

EDSREP 009 T 01 G 

Protocol: BCX4430-106-DMID18-0013


# 10.2 Pharmacokinetic Population

The PK population will include all subjects for whom at least 1 PK parameter can be estimated. The PK population will be the primary population for the PK analysis.

# 11.0 Subject Disposition

The number and percentage of subjects in each analysis population, who complete as well as withdraw from the study prematurely, and a breakdown of the corresponding reasons for withdrawal will be presented for the safety population. A listing of screened subjects and reasons for screen failure will also be presented.

# 12.0 Protocol Deviations

Important protocol deviations/violations will be listed as well as included in the CSR.

# 13.0 Demographic and Baseline Characteristics

# 13.1 Demographics

Subject demographics will be summarized descriptively for all subjects by cohort. The summary will include the subjects' age (in years), sex, race, ethnicity, weight (kg), height (cm), and body mass index (BMI) (in kg/m²). Demographic characteristics will be summarized for the safety and PK populations.

All demographic data, as collected during the screening visit, will be listed by subject.

# 13.2 Medical History

Medical history will be categorized by preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) Version 21.1 and will be listed by subject.

# 13.3 Screening Results

All screening results (including eligibility criteria) will be listed by subject.

### 14.0 Prior and Concomitant Medications

Prior and concomitant medications will be categorized by medication group and subgroup according to the World Health Organization (WHO) Drug Dictionary Version September 2018 and listed by subject. Medications with an end date prior to the first dose of study drug will be considered prior medications and will be identified in the listing. Concomitant medications will include records with a start date on the same date or after the first study drug administration, and records with a start date before the date of first study medication that are indicated as ongoing. If a partial date allows a medication to be considered concomitant it will be categorized as such. Records without a start date are assumed to have started before the date of first study drug administration. Records without an end date are assumed to be ongoing.

# 15.0 Treatment Exposure

The number of subjects who receive study drug will be summarized by cohort and treatment for the safety population. All study drug administration data (including meal data indicating fasting status) will be listed by subject.

Pharmacokinetic Analyses

EDSREP 009 T 01 G 



# 16.0 Pharmacokinetic Variables

# 16.1.1 Plasma Variables

- Plasma concentrations of galidesivir.
- Plasma PK parameters of galidesivir.

Venous blood samples will be collected to determine the plasma concentrations of BCX4430. The plasma concentration summaries and figures with mean values described in this section will be created using the safety population. The plasma PK parameter summaries and statistical analyses described in this section will be created using the PK population.

| Plasma PK Pa | rameters | |
|---|---|---|
| Parameter | Description | Programming Notes |
| | | AUCINF_obs from WNL |
| AUCinf | Area under the concentration versus time curve extrapolated to infinite time, calculated as AUC <sub>last</sub> + $(C_{last}/\lambda_z)$ | If valid lambda_z is not present, then parameter is flagged in listings and will not be used in summary statistics. |
| | | AUClast from WinNonlin |
| AUCt | Area under the concentration versus time curve from time zero to time "t"; may be denoted as AUC <sub>last</sub> if the "t" is the last timepoint with a measurable concentration | If actual time deviates >20% from nominal time, then AUC <sub>1</sub> will be flagged in listings and will not be used in statistical analyses. If valid λ <sub>z</sub> is not present, then AUC <sub>1</sub> is flagged in listings and will not be used in statistical analyses. |
| | | AUC_%Extrap_obs from WinNonlin |
| % AUC <sub>exp</sub> | Percentage of AUC extrapolated between AUC <sub>last</sub> and AUC <sub>inf</sub> | Listed only |
| | | Clast from WinNonlin |
| C <sub>last</sub> | Last measurable concentration of drug | If actual time at T <sub>last</sub> deviates >20% from nominal time, then parameter is flagged in listings and will not be used in summary statistics. |
| | | Tlast from WinNonlin |
| T <sub>last</sub> | Time of last measurable concentration of drug | If actual time at T <sub>last</sub> deviates >20% from nominal time, then parameter is flagged in listings and will not be used in summary statistics |
| C <sub>max</sub> | Maximum observed concentration of drug | C <sub>max</sub> from WinNonlin |



| Plasma PK Parameters | | |
|---|---|---|
| Parameter | Description | Programming Notes |
| | | HL_Lambda_z from<br>WinNonlin |
| t <sub>1/2</sub> | Estimate of the terminal elimination half-life of the drug | If valid $\lambda_z$ is not present, then parameter is flagged in listings and will not be used in summary statistics. |
| CL | CL = Dose/AUC where "Dose" is the dose of the drug and AUC = AUC <sub>inf</sub> | CL_obs from WinNonlin |
| | | Lambda_z from WinNonlin |
| $\lambda_{z}$ | Terminal elimination rate constant, estimate by linear regression of the terminal elimination phase of the concentration of drug versus time curve | If Rsq < 0.80 then parameter is flagged in listings and will not be used in summary statistics. |
| | Volume of distribution of the drug | Vz_obs from WinNonlin If valid $\lambda_z$ is not present, then parameter is flagged in listings and will not be used in summary statistics. |
| Vz | volume of distribution of the drug | Tmax from WinNonlin |
| T <sub>max</sub> | Time to C <sub>max</sub> | I max nom vviimomili |

Note: In all derivations of PK parameters, BQL values at the beginning of the profile will be set to zero, whereas BQL values that occur after the first quantifiable point will be considered missing. Samples that are BQL but are between two samples with detectable concentrations will be excluded from PK analysis.

# 16.1.2 Urine Variables

- Urine concentrations of galidesivir.
- Urine PK parameters of galidesivir.

Urine samples will be collected to determine the concentrations of galidesivir. The urine PK parameter summaries described in this section will be created using the PK population.

| Urine PK Parameters | | |
|---|---|---|
| Parameter | Description | Programming Notes |
| Ct1-t2 | Concentration (of the unchanged drug) in the collection interval t1-t2. | Directly from data, no calculation required. |
| Vt1-t2 | Volume of the urine collected in the interval t1-t2 | Measured in the clinic, captured on the CRF, no calculation required. |

EDSREP 009 T 01 G 





| Urine PK Parameters | | |
|---|---|---|
| Parameter | Description | Programming Notes |
| | Amount of drug excreted unchanged into urine in the interval t1-t2, calculated as the urine volume times the urine concentration for each interval. | Ct1-t2 *Vt1-t2 |
| Aet1-t2 | Intervals: 0-12 h, 12-24 h, 24-48 h, 48-72 h, 72-96 h, 0-96h (cumulative) | |
| % Doseexcreted,t1-t2 | Percentage of given dose excreted in the urine as unchanged drug Intervals: 0-12 h, 12-24 h, 24-48 h, 48-72 h, 72-96 h, 0-96h (cumulative) | Aet1-t2/Dose*100 Dose will be converted to match units of Ae |
| | | CLr=Ae0-t1/AUC0-t1 CLr parameter will be |
| $CL_{f}$ | Renal clearance of unchanged drug cumulatively over all collection intervals | calculated according to time matched AUC. |

Note: Urine PK parameters will be estimated in SAS based on the recorded urine concentrations and volumes. In estimating the parameters, all missing values will be recorded as missing and all BLQ values will be set to zero. If a missing value is encountered, the cumulative parameters will not be calculated for that subject.

#### 16.2 Pharmacokinetic Summaries

# 16.2.1 Plasma Concentrations

Plasma concentrations for BCX4430 below the quantifiable limit (BQL) will be set to zero in the computation of mean concentration values. Descriptive statistics including n, arithmetic mean, SD, arithmetic CV%, geometric mean, geometric CV%, geometric n (the number of subjects with an observation who were included in the natural logarithmic transformation) median, min, and max will be used to summarize the plasma concentrations by treatment at each scheduled time point. If more than half of the subjects in a given cell have values BQL, then the descriptive statistics will not be presented and will instead display as BQL for the mean and minimum. Except for n and maximum, all other statistics will be missing. Any value less than BQL will be presented as BQL.

Linear and semi-logarithmic plots of the arithmetic mean and median plasma concentrations by scheduled sampling time will be provided by treatment. These plots will show time in hours. The plots will match the summary table results and will not have an observation at a given time point if more than half of the subjects have values BQL. Mean plots will include SD error bars when plotted on a linear scale and log scale.

Linear and semi-logarithmic plots of the individual plasma concentrations by actual sampling time will be provided by subject (1 subject per page). These plots will show time in hours. Individual plots will use the BQL handling procedure described below for "Plasma Pharmacokinetic Parameters".

All individual subject plasma concentration data will be listed by cohort and treatment.

#### 16.2.2 Plasma Pharmacokinetic Parameters

Plasma PK parameters for BCX4430 will be estimated using non-compartmental methods with WinNonlin®.

The plasma PK parameters will be estimated from the concentration-time profiles. In estimating the PK parameters. BQL values at the beginning of the profile will be set to zero. BQL values that occur after the first quantifiable point will be considered missing. Samples that are BQL but are between two samples with detectable concentrations will be excluded from PK analysis.

EDSREP 009 T 01 G 



Actual sampling times, rather than scheduled sampling times, will be used in all computations involving sampling times. If the actual time or dose time is missing, the scheduled time may be substituted in order to calculate the PK parameter.

Determination of points to be included in  $\lambda_z$  range will follow the Guideline for Defining, Calculating and Summarizing Pharmacokinetic / Pharmacodynamic Parameters (EDSREP 009 R 01) and rule will be noted in table and listing footnotes.

Descriptive statistics (n, arithmetic mean, SD, arithmetic CV%, geometric mean, geometric CV%, median, min, and max) will be used to summarize the calculated PK parameters by treatment. For  $T_{max}$ ,  $T_{lag}$ , and  $T_{last}$ , only n, median, min, and max will be presented.

Individual PK parameters AUCt, AUCinf, and Cmax with corresponding geometric means will be shown graphically for each treatment.

All individual subject PK parameters will be listed by treatment and period.

### 16.2.3 Urine Pharmacokinetic Parameters

Urine PK parameters will be estimated in SAS based on the recorded urine concentrations and volumes. In estimating the parameters, all missing values will be recorded as missing and all BLQ values will be set to zero. If a missing value is encountered, the cumulative parameters will not be calculated for that subject. Summaries of amounts excreted by treatment and scheduled collection interval (Aet1-t2), including cumulative amount excreted, fraction excreted by treatment and scheduled collection interval (% Dose<sub>excreted,t1-t2</sub>), including cumulative fraction excreted, and renal clearance (CLr) will be provided. Descriptive statistics (n, arithmetic mean, SD, arithmetic CV%, geometric mean, geometric CV%, median, min, and max) will be used to summarize the calculated PK parameters by treatment.

## 16.2.4 Dose Proportionality Analyses

#### 16.2.4.1 Power Model

The assessment of dose proportionality for the PK parameters of BCX4430 will use a power model approach (including all doses). A model with In-transformed dose (dose continuous) as a fixed effect and subject as a random effect will be applied to the following In-transformed PK parameters: AUCt, AUCinf, and Cmax. Although there is no formal statistical hypothesis tested for this secondary objective, there will be evidence for dose-proportionality for each PK parameter if the 90% confidence interval (CI) of the fixed slope for In-dose contains 1. No adjustment for multiplicity will be performed for the set 3 of PK parameters.

The SAS pseudo code for the power model is as follows:

```
data adpp;
set adpp;
in_auc = log(auc);
In_dose = log(dose);
run;

proc mixed data=adpp method=reml;
by parameter;
class subject;
model in_auc = In_dose / ddfm=kr cl alpha=0.1;
random subject;
run;
```

#### 16.2.4.2 ANOVA Model Pairwise Comparisons

Following log-e transformation, dose-normalized PK parameters will be analyzed with an ANOVA model using PROC MIXED. Each dose will be compared with a reference dose on a pair-wise basis. Pairwise

EDSREP 009 T 01 G 




Protocol: BCX4430-106-DMID18-0013 Version Date: 10-April-2019

comparisons of the ratio of GLS means and the corresponding 90% CI will be estimated for each PK parameter of interest. Although there is no formal statistical hypothesis tested for this secondary objective, if the 90% CI for the geometric LSM ratio falls completely within the 0.8 to 1.25 equivalence region then dose proportionality is indicated for the specific comparison. No adjustment for multiplicity will be performed for the set of descriptive pairwise comparisons.

The SAS PROC MIXED pseudo code for the pairwise comparison for the ANOVA model is as follows:

```
data adpp;
set adpp;
In_auc_dose = log(auc)/dose;
run;
ods output diffs=diffs;
ods output lsmeans=lsmeans;
proc mixed data=adpp method=reml;
by parameter;
class dose;
model In_auc_dose = dose / ddfm=kr;
Ismeans dose / pdiff alpha=0.1 cl;
run;
```

# 17.0 Safety Analyses

The safety summaries described in this section will be created using the safety analysis population. Safety analyses will be performed separately for each cohort.

# 17.1 Safety Variables

The following safety variables will be included:

- Adverse events
- Clinical laboratory evaluations
  - Cardiac markers (troponin and creatine kinase-MB [CK-MB])
  - Chemistry
  - Coagulation
  - Hematology
  - Urinalysis
  - Serology
  - Pregnancy
  - Alcohol breath test and urine drug screen
- Vital signs
  - Systolic blood pressure
  - o Diastolic blood pressure
  - Pulse rate
  - Oral body temperature
- Electrocardiograms
  - Heart rate
  - o RR interval
  - o PR interval
  - QRS duration
  - QT interval
  - QT interval corrected using Fredericia's method (QTcF)
- Physical examination findings


#### 17.1.1 Adverse Events

An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant that does not necessarily have a causal relationship with treatment. TEAEs are those which occur during or after the administration of the first dose of study drug. All TEAE summaries will be presented alphabetically by system organ class, with preferred terms sorted in decreasing order of frequency within each system organ class based on MedDRA Version 21.1.

The following missing data will be imputed (for calculations only) as defined:

- Missing AE start and / or end times for the calculation of onset and duration will be assumed to be at 00:01 for a start time and 23:59 for end times
- Missing AE severity or relationship will be assumed to be severe or related, respectively
- Missing AE start times for the determination of treatment emergence will be assumed to occur after treatment unless partial date documents the AE as happening prior to treatment
- Missing AE start times for the determination of treatment assignment will be assumed to occur after treatment on the recorded date 1 minute after dosing
- Missing AE start date will be assumed to be after treatment for the determination of TEAE but will
  not be attributed to a specific study drug

A summary of the number and percentage of subjects reporting AEs, TEAEs, serious AEs (SAEs), and who discontinue study drug due to an AE will be provided by cohort and overall for the study.

A summary of the number and percentage of subjects reporting each TEAE will be provided by cohort and treatment, and overall. Counting will be done by subject, not by event; subjects will only be counted once within each system organ class or preferred term.

A summary of the number and percentage of subjects reporting each TEAE will be provided by relationship to treatment (BCX4430 formulation, as recorded on eCRF) and by cohort and treatment, and overall. Subjects with multiple events will be counted under the category of their most-related event within each system organ class or preferred term.

A summary of the number and percentage of subjects reporting each TEAE will be provided by severity (as recorded on eCRF) and by cohort and treatment, and overall within each cohort. Subjects with multiple events will be counted under the category of their most severe event within each system organ class or preferred term.

All AEs (including non-treatment-emergent AEs) recorded on the eCRF will be listed by subject.

A separate listing of AEs leading to study drug discontinuation will be provided by subject.

### 17.1.2 Deaths and Serious Adverse Events

A listing of deaths and a listing of SAEs will be provided by subject.

#### 17.1.3 Laboratory Data

Clinical laboratory data will be presented using units from the study data tabulation model (SDTM) Controlled Terminology.

A descriptive statistics summary of continuous laboratory results and derived changes from baseline for cardiac markers, chemistry, coagulation, hematology, and urinalysis will be provided by cohort and scheduled timepoint.

Laboratory abnormalities outside of the normal laboratory reference ranges and associated grades (according to study specific DMID criteria specified in the 2014 DMID Adult Toxicity Grading Scale in Appendix 5) should be denoted where possible. For those analyte results that are out of the normal range and do not have an established DMID toxicity criteria, the severity grading will be provided by the PI. The number and percentage of subjects experiencing treatment-emergent graded toxicities will be summarized.

FDSRFP 009 T 01 G 


A shift table describing the change in continuous clinical laboratory values from baseline to follow-up (number and percentage of subjects) will also be provided. The following categories will be used: Normal, DMID Grade 1, DMID Grade 2, DMID Grade 3, DMID Grade 4.

All laboratory data will be listed by subject, including laboratory variables not listed in the protocol.

A separate listing of out-of-range values will also be provided. Normal ranges will be used directly from the clinical laboratory and will be included in the listings for reference. Flags for high and low values will be provided in the listings.

# 17.1.4 Vital Signs

A descriptive statistics summary of vital signs and derived changes from baseline will be provided by cohort and treatment, and scheduled timepoint. Baseline is defined as measurement prior to initiation of treatment on Day 1 of each treatment period, where available.

All vital signs data will be listed by subject.

# 17.1.5 Electrocardiograms

A descriptive statistics summary of 12-lead ECG parameters and derived changes from baseline will be provided by cohort and treatment, and scheduled timepoint. Where triplicate ECGs are taken, the average parameter values of the triplicates will be reported. Baseline is defined as the average of triplicate measurements prior to initiation of treatment on Day 1 of each treatment period, where available.

A summary table for QTcF categories (<=450 msec, >450 to <= 480 msec, >480 to <=500 msec, and > 500 msec) by cohort and treatment, and timepoint will be presented. The table will also summarize the number and percentage of subjects with change from baseline for categories of <= 30 msec, 30 msec to <= 60 msec, and > 60 msec.

All 12-lead ECG parameters, physician's conclusions, and corresponding abnormalities and will be listed by subject.

Descriptive statistics will be provided to summarize mean ECG parameters (observed and changes from baseline) by treatment, visit, and scheduled time.

### 17.1.6 Cardiac Telemetry

A listing of the cardiac telemetry data will include the start and stop times of telemetric observation, the occurrence of any arrythmia or tachycardia of Grade 2 or higher (i.e. heart rate greater than 115 beats per minute), and the clinical evaluation of clinical significance of any arrythmia or tachycardia.

#### 17.1.7 Echocardiograms

A listing of the echocardiogram data will include the date and time of the assessment, the ejection fraction, and any clinical finding confirmed by cardiologist.

# 17.1.8 Physical Examination

All physical examination data will be listed by subject.

EDSREP 009 T 01 G 


# References

SAS Institute, Inc., SAS® Version 9.4 software, Cary, NC.

Clinical Study Protocol. A Phase 1 Drug Interaction Study to Evaluate the Effect of BCX4430 on the Pharmacokinetics of Danazol, Amlodipine and Desipramine in Healthy Subjects. Version 1.0, Final, 07 Mar 2018.

Gough K, Hutchison M, Keene O, Byrom B, Ellis S, Lacey L, McKellar J. (1995). Assessment of dose proportionality: Report from the statisticians in the pharmaceutical industry / pharmacokinetics UK joint working party, Drug Information Journal, Vol. 29:1039-1048.

Patroneva A, Connolly SM, Fatato P, et al. (2008). An assessment of drug-drug interactions: the effect of desvenlafaxine and duloxetine on the pharmacokinetics of the CYP2D6 probe desipramine in healthy subjects. Drug Metab Dispos 36(12): 2484-2491.

Vincent J, Harris SI, Foulds G, et al. (2000). Lack of effect of grapefruit juice on the pharmacokinetics and pharmacodynamics of amlodipine. Br J Clin Pharmacol 50(5): 455-463.

EDSREP 009 T 01 G 

Protocol: BCX4430-106-DMID18-0013 Version Date: 10-April-2019

# **Appendix 1: Glossary of Abbreviations**

# Glossary of Abbreviations:

AE Adverse event

ADaM Analysis data model

AUC Area under the concentration-time curve

AUC<sub>inf</sub> Area under the concentration versus time curve extrapolated to infinite time

AUCt Area under the concentration time curve from time 0 to time t (hours)

AUC%extrap Percentage of AUC extrapolated between AUCt and AUCinf.

BQL Below the quantifiable limit

Cl Confidence interval

C<sub>last</sub>
Concentration observed at the last quantifiable time point.

CL/F
Apparent oral clearance after administration of the drug

C<sub>max</sub> Maximum plasma concentration.

CSR Clinical study report
CRU Clinical research unit
CV Coefficient of variation

DMID Division of Microbiology and Infectious Disease

ECG Electrocardiogram

eCRF Electronic case report form
EDS Early Development Services

LSM Least squares means

Max Maximum

MedDRA Medical Dictionary for Regulatory Activities

Min Minimum

PK Pharmacokinetic
QC'd Quality controlled

SAP Statistical analysis plan
SAE Serious adverse event

SD Standard deviation

TEAE Treatment-emergent adverse event

TFL(s) Tables, figures and listings

T<sub>lag</sub> Elapsed time from dosing at which analyte was first quantifiable in a

concentration vs. time profile

 $T_{last}$  Time of  $C_{last}$   $T_{max}$  Time of  $C_{max}$ 

Protocol: BCX4430-106-DMID18-0013 Version Date: 10-April-2019

| T <sub>1/2</sub> | Terminal phase half-life expressed in time units |
|------------------|--------------------------------------------------|
| Vz/F | Apparent volume of distribution of the drug. |
| WHO | World Health Organization |
| $\lambda_z$ | Terminal elimination rate constant |



Appendix 2: Schedules of Assessments from Protocol

# **Schedule of Assessments**

| Assessment | Screening | CRU | | | | | Return to<br>CRU for PK<br>Sample | Follow-up or<br>Early<br>Termination<br>Visit | |
|---|---|---|---|---|---|---|---|---|---|
| | Day -28<br>to -2 | Day ~1<br>(Admission) | Day 1<br>Baseline<br>(Pre-<br>dose) | Day 1<br>(Post<br>dose) | Day 2 | Day 3 | Day 4<br>(Discharge) | Day 5, Day 7,<br>Day 14 <sup>n</sup> | Day 21 + 2 |
| Informed consent | X | | | | | | | | |
| Inclusion/exclusion criteria | X | Х | | | | | | | |
| Medical history | X | X | | | | | | | |
| Weight/height/BMI | X | Xa | | | | | | | |
| Drugs of abuse<br>screen/urine alcohol<br>test/urine cotimine<br>screen | X | Х | | | | | | | |
| HIV/HCV/HBV<br>serology | Х | | | | | | | | |
| Physical<br>examination <sup>b</sup> | Х | X | Х | Х | X | X | X | | х |
| Concomitant medications | Х | X | X | X | Х | X | X | X | х |
| ECG | Χ¢ | | Xc | Xď | Xd | Xd | X <sup>d</sup> | | X <sup>d</sup> |
| Cardiac telemetry | | | Xe | Xe | | | | | |

EDSREP 009 T 01 G 

Protocol: BCX4430-106-DMID18-0013


| Assessment | Screening | In Clinic (CRU) Study Period | | | | | Return to<br>CRU for PK<br>Sample | Follow-up or<br>Early<br>Termination<br>Visit | |
|---|---|---|---|---|---|---|---|---|---|
| | Day -28<br>to -2 | Day -1<br>(Admission) | Day 1 Baseline (Pre- dose) | Day 1<br>(Post<br>dose) | Day 2 | Day 3 | Day 4<br>(Discharge) | Day 5, Day 7,<br>Day 14 <sup>n</sup> | Day 21 + 2 |
| ECHO <sup>f</sup> | | $X^{f}$ | | | | Xf | | | |
| Vital signs | X | X | Xg | Xg | Xg | X | X | | X |
| Pregnancy testh | X | X | | | | | | | X |
| FSH <sup>i</sup> | X | | | | | | | | |
| Clinical chemistry/<br>hematology | Х | X <sup>m</sup> | | X | X | X | X | | Х |
| Urinalysis | X | X <sup>m</sup> | | | X | X | X | | X |
| aPTT/PT | X | X <sup>m</sup> | | | | | X | | X |
| Testosterone | | X <sup>m</sup> | | | | | X | | X |
| Troponin I | | X <sup>m</sup> | | | | | X | | X |
| CK-MB | | Xm | | | | | X | | X |
| Cystatin C and<br>NGAL | | X <sup>m</sup> | | 3 | | | X | | X |
| UACR | X | Xm | | | | | X | | X |
| Plasma for galidesivir<br>PK analysis <sup>k</sup> | | | X <sup>k</sup> | X <sup>k</sup> | X | X | X | X | X |
| Urine for galidesivir<br>PK analysis <sup>1</sup> | | | X | X | X | X | X | | |
| AE assessment | | X | X | X | X | X | X | X | X |
| Study drug dosing | | | | Х | | | | | |

Protocol: BCX4430-106-DMID18-0013


Abbreviations: AE = adverse event; aPTT = activated partial thromboplastin time; BMI = body mass index; CK-MB = creatine kinase-MB; CRU = clinical research unit; ECG = electrocardiogram; ECHO = echocardiogram; FSH = follicle-stimulating hormone; HBV = hepatitis B virus; HCV = hepatitis C virus; HIV = human immunodeficiency virus; NGAL = neutrophil gelatinase-associate lipocalin; PK = pharmacokinetic; PT = prothrombin time; UACR = urine albumin-to-creatinine ratio.

- a. Weight only.
- b. A physical examination consisting of the head and neck, skin, chest (lungs and heart), abdoinen (gastrointestinal tract, liver, spleen and kidneys), back, musculoskeletal system, and neurologic system should be conducted at screening and on Day 4 prior to discharge. Breast and genitourinary system do not require examination unless the potential subject indicates a complaint or comorbidity that could result in exclusion. All other physical exams will be symptom directed. The site of infusion should be checked for any changes in skin.
- c. Three (3) serial ECGs will be performed at screening and baseline 1–3 minutes apart. Pre-dose ECG should be collected within ≤ 2 hours of the first dose.
- d. 12-lead ECGs will be conducted on Day 1 at 2 and 4 hours post dose (post start of the infusion) and on Day 2 at 24 hours post dose. An acceptable window is ± 10 minutes from the nominal time point. All subsequent ECGs are daily.
- e. Cardiac telemetry will be initiated ≥ 2 hours prior to administration of the dose and will continue for 24 hours after the infusion is started. Subjects may be disconnected for bathroom, hygiene needs, and for 20-minute periods 3 times a day for meals. In addition, subjects may be disconnected for 10 minutes every 2 hours while awake for mild physical exercise such as walking or calf exercises.
- f. The ECHO may be performed at any time from screening to Day -1 for eligibility determination. An ECHO should also be performed on Day 3. An acceptable window for the Day 3 ECHO is up until Day 4 discharge.
- g. Vital signs (except temperature) will be obtained pre-dose (within 2 hours of dosing) 1, 2, 4, and 8 hours post dose (post start of the infusion) on Day 1, at 24 hours post dose on Day 2 and once per day where indicated. Oral temperature will be obtained at 8 hours post dose on Day 1 and at 24 hours post dose on Day 2. Subjects should be rested for 10 minutes in the supine position prior to vital sign measurements.
- h. A serum pregnancy test will be administered at screening to all women; all other pregnancy tests performed during the study may be urine pregnancy tests.
- i. An FSH level will be measured in women who report that they have been postmenopausal  $\leq 2$  years.
- j. Free testosterone will be measured in male subjects.
- k. Plasma for PK galidesivir analysis will be collected pre-dose, 30 min (halfway through the infusion), 1 h (end of the infusion), 1.25 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 36 h, 48 h, 60 h, 72 h, and 96 h following the start of the infusion. The pre-dose PK sample must be collected within ≤ 1 hour of the dose. Assessment windows around each PK draw will be ± 2 minutes for sampling times up to 2-hour post dose and from 2-hour post dose onward, ± 10 minutes while subject is confined in the unit. All sample times are from the start of the infusion.
- 1. For the analysis of urinary excretion of galidesivir, an aliquot of urine will be collected pre-dose (0 hour) and all urine will be collected for the following post dose intervals: 0-12 hours, 12-24 hours, 24-48 hours, 48-72 hours, and 72-96 hours. All sample times are from the start of the infusion.
- m. Baseline for study post dose comparisons. NGAL, cystatin C, UACR, testosterone, troponin l, and CK-MB can be collected on Day -1 or Day 1 (pre-dose).
- n. Subjects will return to the CRU to have a plasma PK sample collected on Day 5 (+1), Day 7 (+1), and Day 14 (±1). This visit is intended to be a short visit (approximately 1-2 hours) and can take place at any time during the specified window. A plasma PK sample will also be collected at the follow-up visit on Day 21.

# Appendix 3: List of End of Text Outputs

| | Text Tables and Figures: | T |
|---|---|---|
| Output | Title | Analysis Population |
| Section 14.1 – D | isposition and Demographic Data | |
| Table 14.1.1 | Summary of Subject Disposition | All Subjects |
| Table 14.1.2.1 | Summary of Demographics | Safety |
| Table 14.1.2.2 | Summary of Demographics | PK |
| Table 14.1.3 | Summary of Study Drug Administration | Safety |
| Section 14.2 – P | lasma Pharmacokinetic Data | |
| Table 14.2.1 | Summary of BCX4430 Plasma Concentrations | Safety |
| Table 14.2.2 | Summary of BCX4430 Plasma Pharmacokinetic Parameters | PK |
| Table 14.2.3 | Summary of BCX4430 Urine Pharmacokinetic Parameters | PK |
| Table 14.2.3.1 | Statistical Analysis of the Dose Proportionality: Power Model | PK |
| Table 14.2.3.2 | Statistical Analysis of the Dose Proportionality: ANOVA Model of<br>Pairwise Comparisons | PK |
| Figure 14.2.4 | Plot of Mean (±SD) BCX4430 Plasma Concentrations vs Time on a Linear Scale | Safety |
| Figure 14.2.5 | Plot of Mean BCX4430 Plasma Concentrations vs Time on a Semi-Log Scale | Safety |
| Figure 14.2.6 | Plot of Median BCX4430 Plasma Concentrations vs Time on a Linear Scale | Safety |
| Figure 14.2.7 | Plot of Individual BCX4430 Plasma Concentrations vs Time on a Linear Scale | Safety |
| Figure 14.2.8 | Plot of Individual BCX4430 Plasma Concentrations vs Time on a Semi-<br>Log Scale | Safety |
| Figure 14.2.9 | Scatter Plot of Individual BCX4430 Plasma Pharmacokinetic Parameters | PK |
| Section 14.3 – S | afety Data | |
| Table 14.3.1.1 | Summary of Adverse Events | Safety |
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term | Safety |
| Table 14.3.1.3 | Summary of Treatment Emergent Adverse Events by Relationship to BCX4430 | Safety |
| Table 14.3.1.4 | Summary of Treatment Emergent Adverse Events by Severity | Safety |
| Table 14.3.2 | Listing of Serious Adverse Events | All Subjects |
| Table 14.3.3 | Listing of Deaths | All Subjects |
| Table 14.3.4 | Listing of Abnormal Laboratory Values | All Subjects |
| Table 14.3.5.1 | Summary of Laboratory Results | Safety |
| Table 14.3.5.2 | Summary of Laboratory Shifts from Baseline | Safety |

EDSREP 009 T 01 G 

| Table 14.3.5.3 | Summary of Treatment Emergent Graded Laboratory Toxicities | Safety |
|---|---|---|
| Table 14.3.6 | Summary of Vital Signs | Safety |
| Table 14.3.7.1 | Summary of 12-Lead Electrocardiogram Results | Safety |
| Table 14.3.7.2 | Summary of QTcF Categorical Findings | Safety |

| | Text Listings:<br>T ـ | |
|---|---|---|
| Output | Title | |
| Section 16.2.1 – | Disposition | |
| Listing 16.2.1.1 | Subject Disposition | |
| Listing 16.2.1.2 | Eligibility Criteria | |
| Section 16.2.2 – | Protocol Deviations | |
| isting 16.2.2 | Important Protocol Deviations | |
| Section 16.2.3 - | Excluded Subjects | |
| _isting 16.2.3 | Analysis Populations | |
| Section 16.2.4 - | Demographics and Baseline Characteristics | |
| _isting 16.2.4.1 | Subject Demographics | |
| Listing 16.2.4.2 | Medical History | |
| isting 16.2.4.3 | Prior and Concomitant Medications | As any artifact they first |
| Section 16.2.5 - | Compliance | |
| isting 16.2.5.1 | Study Drug Administration | |
| isting 16.2.5.2 | Meal Administration | |
| Section 16.2.6 - | Response Data | |
| _isting 16.2.6.1 | Plasma Concentrations | |
| _isting 16.2.6.2 | Plasma Pharmacokinetic Parameters | . 10 |
| isting 16.2.6.3 | Urine Pharmacokinetic Parameters | |
| Section 16.2.7 - | Adverse Events Data | |
| _isting 16.2.7.1 | Adverse Events | |
| isting 16.2.7.2 | Adverse Events Leading to Study Drug Discontinuation | |
| Section 16.2.8 - | Laboratory Data | |
| _isting 16.2.8.1 | Clinical Laboratory Results - Cardiac Markers | |
| _isting 16.2.8.2 | Clinical Laboratory Results – Chemistry | |
| isting 16.2.8.3 | Clinical Laboratory Results – Coagulation | |
| _isting 16.2.8.4 | Clinical Laboratory Results – Hematology | |
| isting 16.2.8.5 | Clinical Laboratory Results – Urinalysis | |
| Listing 16.2.8.6 | Clinical Laboratory Results – Serology | |
| _isting 16.2.8.7 | Clinical Laboratory Results – Pregnancy and FSH | |
| Listing 16.2.8.8 | Clinical Laboratory Results - Urine Drug and Alcohol Screen | |

EDSREP 009 T 01 G 

| Listing 16.2.9 | Vital Signs |
|-----------------|-----------------------------------|
| Listing 16.2.10 | 12-Lead Electrocardiogram Results |
| Listing 16.2.11 | Cardiac Telemetry Results |
| Listing 16.2.12 | Echocardiogram Results |
| Listing 16.2.13 | Physical Examination Findings |

| Other Appendix | Outputs: |
|----------------|----------|
| Output | Title |

Appendix 16.1.9.2 Statistical Appendices

# Appendix 4: Shells for Post-Text Tables, Figures and Listings Shells are provided in a separate document.

| Clinical Adverse<br>Events | | | |
|---|---|---|---|
| VITAL SIGNS | Mild<br>(Grade 1) | Moderate (Grade 2) | Severe<br>(Grade 3) |
| Fever (°C) ** | 38.0 – 38.4 | 38.5 – 38.9 | ≥39.0 |
| (°F) ** | 100.4 – 101.1 | 101.2 – 102.0 | >102.0 |
| ** Oral temperature;<br>either °C or °F for inc | | verages or smoking. A pro | otocol should select |
| Tachycardia - beats<br>per minute | 101 – 115 | 116 – 130 | > 130 or ventricular<br>dysrhythmias |
| Bradycardia - beats<br>per minute | 50 – 54 or 45-50<br>bpm if baseline <60<br>bpm | 45 – 49 or 40-44 if baseline <60bpm | < 45 or <40bpm if baseline <60bpm |
| Hypertension#<br>(systolic)- mm Hg | 141-150 | 151-160 | > 160 |
| Hypertension#<br>(diastolic) - mm Hg | 91-95 | 96-100 | > 100 |

| Hypotension<br>(systolic) - mm Hg | 85-89 | 80-84 | < 80 |
|---|---|---|---|
| Tachypnea – | 23-25 | 26-30 | >30 |
| breaths per minute | | | |
| CARDIOVASCULA<br>R | Grade 1 | Grade 2 | Grade 3 |
| Arrhythmia | | asymptomatic,<br>transient signs, no Rx<br>required | recurrent/persistent;<br>symptomatic Rx<br>required |
| QTcF interval prolonged (msec) | Asymptomatic, QTcF<br>>450-480 msec | Asymptomatic, QTcF<br>>480-500 msec OR<br>increase in interval 30-<br>60 msec from baseline | Asymptomatic, QTcF<br>>500 msec OR<br>increase in interval<br>>60 msec from<br>baseline |
| Hemorrhage, Blood<br>Loss | Estimated blood loss < 100 mL | Estimated blood loss > 100 mL, no transfusion required | Transfusion required |
| RESPIRATORY | Grade 1 | Grade 2 | Grade 3 |
| Cough | Transient- no treatment | Persistent cough; | Interferes with daily activities |
| Bronchospasm,<br>Acute | transient; no<br>treatment; 71% -<br>80% FEV1 of peak<br>flow | requires treatment;<br>normalizes with<br>bronchodilator; FEV1<br>60% - 70% (of peak<br>flow) | no normalization with<br>bronchodilator; FEV1<br><60% of peak flow |
| Dyspnea | Does not interfere with usual and social activities | Interferes with usual<br>and social activities, no<br>treatment | Prevents daily and usual social activity or requires treatment |
| GASTROINTESTIN<br>AL | Grade 1 | Grade 2 | Grade 3 |
| Nausea | No interference with activity | Some interference with activity | Prevents daily activities |
| Vomiting | No interference with activity or 1 - 2 episodes/24 hours | Some interference with activity or > 2 episodes/24 hours | Prevents daily activity or requires IV hydration |

| Iliness or clinical<br>adverse event (as<br>defined according to<br>applicable<br>regulations) | Transient or mild symptoms; no limitation in activity; no intervention required. The AE does not interfere with the participant's normal functioning level. It may be an annoyance. | Symptom results in mild to moderate limitation in activity; no or minimal intervention required. The AE produces some impairment of functioning, but it is not hazardous to health. It is uncomfortable or an embarrassment. | Symptom results in significant limitation in activity; medical intervention may be required. The AE produces significant impairment of functioning or incapacitation. |
|---|---|---|---|
| All Other conditions | Mild<br>(Grade 1) | Moderate (Grade 2) | Severe<br>(Grade 3) |
| Myalgia | No interference with activity | Some interference with activity | Significant; prevents daily activity |
| Fatigue | No interference with activity | Some interference with activity | Significant; prevents daily activity |
| Headache | No interference with activity | Repeated use of non-<br>narcotic pain reliever ><br>24 hours or some<br>interference with<br>activity | Significant; any use of narcotic pain reliever or prevents daily activity |
| Allergic<br>Reaction/Hypersens<br>itivity | pruritus without rash | localized urticaria | generalized urticaria;<br>angioedema or<br>anaphylaxis |
| SYSTEMIC | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
| Diarrhea | 2 - 3 loose or watery<br>stools or < 400<br>gms/24 hours | 4 - 5 loose or watery<br>stools or 400 - 800<br>gms/24 hours | 6 or more loose or<br>watery stools or ><br>800gms/24 hours or<br>requires IV hydration |

EDSREP 009 T 01 G 

| Laboratory Adverse<br>Events | | | | | |
|---|---|---|---|---|---|
| Blood, Serum, or Plasma<br>* | Reference | Range ** | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
| Sodium – Hyponatremia<br>mEq/L | 135-146 mr | nol/L | 134 – <lln< td=""><td>132 – 133</td><td>&lt;132</td></lln<> | 132 – 133 | <132 |
| Sodium – Hypernatremia<br>mEq/L | 135-146 mn | nol/L | >ULN - 147 | 148 – 149 | >149 |
| Potassium – Hyperkalemia<br>mEq/L | 3.5-5.3 mm | ol/L | >ULN - 5.4 | 5.5 - 5.6 | >5.6 |
| Potassium – Hypokalemia<br>mEq/L | 3.5-5.3 mm | ol/L | <lln-3.4< td=""><td>&lt;3.4 – 3.3</td><td>&lt;3.3</td></lln-3.4<> | <3.4 – 3.3 | <3.3 |
| Glucose – Hypoglycemia<br>mg/dL | 65-99 mg/d | L | 62 – 64 | 52 – 62 | <52 |
| Glucose – Hyperglycemia<br>Fasting – mg/dL | 65-99 mg/d | L | >ULN - 100 | 101 110 | >110 |
| Glucose – Hyperglycemia<br>Random – mg/dL | 65-139 mg/ | dL | 140 – 159 | 160 – 200 | >200 |
| Blood Urea Nitrogen mg/dL | 7-25 mg/dL | | 26 – 29 | 30 – 34 | >34 |
| Creatinine (Male) - mg/dL | 18Y-19Y | 0.60-1.26<br>mg/dL | >ULN 1.36 | >1.36 – 1.56 | >1.56 |
| | 20Y-49Y | 0.60-1.35<br>mg/dL | >ULN - 1.45 | >1.45 – 1.65 | >1.65 |
| | 50Y-59Y | 0.70-1.33<br>mg/dL | >ULN 1.43 | >1.43 – 1.63 | >1.63 |
| Creatinine (Female)- mg/dL | 18Y-19Y | 0.50-1.00<br>mg/dL | >ULN 1.10 | >1.10 - 1.30 | >1.30 |
| | 20Y-49Y | 0.50-1.10<br>mg/dL | >ULN - 1.20 | >1.20 – 1.40 | >1.40 |
| | 50Y-59Y | 0.50-1.05<br>mg/dL | >ULN 1.15 | >1.15 1.35 | >1.35 |
| Calcium – hypocalcemia<br>mg/dL (Male) | 18Y-19Y | 8.9-10.4<br>mg/dL | 8.8 – <lln< td=""><td>8.3 – 8.7</td><td>&lt;8.3</td></lln<> | 8.3 – 8.7 | <8.3 |
| mg/ac (Male) | 20Y-133Y | 8.6-10.3<br>mg/dL | 8.5 <lln< td=""><td>8.0 – 8.4</td><td>&lt;8.0</td></lln<> | 8.0 – 8.4 | <8.0 |
| Calcium – hypocalcemia<br>mg/dL (Female) | 18Y-19Y | 8.9-10.4<br>mg/dL | 8.8 – <lln< td=""><td>8.3 – 8.7</td><td>&lt;8.3</td></lln<> | 8.3 – 8.7 | <8.3 |
| mg/at (i emale) | 20Y-49Y | 8.6-10.2<br>mg/dL | 8.5 <lln< td=""><td>8.0 – 8.4</td><td>&lt;8.0</td></lln<> | 8.0 – 8.4 | <8.0 |
| | 50Y-133Y | 8.6-10.4<br>mg/dL | 8.5 <lln< td=""><td>8.0 – 8.4</td><td>&lt;8.0</td></lln<> | 8.0 – 8.4 | <8.0 |
| Calcium – hypercalcemia<br>mg/dL (Male) | 18Y-19Y | 8.9-10.4<br>mg/dL | >ULN - 10.5 | 10.6 – 11.0 | >11.0 |
| marar (mais) | 20Y-133Y | 8.6-10.3<br>mg/dL | >ULN - 10.4 | 10.5 – 10.9 | >10.9 |
| Calcium – hypercalcemia | 18Y-19Y | 8.9-10.4<br>mg/dL | >ULN - 10.5 | 10.6 10.9 | >10.9 |
| mg/dL (Female) | 20Y-49Y | 8.6-10.2 | >ULN 10.3 | 10.4 – 10.7 | >10.7 |
| | 50Y-133Y | mg/dL<br>8.6-10.4<br>mg/dL | >ULN - 10.5 | 10.6 - 10.9 | >10.9 |

EDSREP 009 T 01 G 

| Magnosium | 1505 | | 40.45 | 144 46 | |
|---|---|---|---|---|---|
| Magnesium – | 1.5-2.5 mg/d | ar. | 1.3 – 1.5 | 1.1 – 1.2 | <1.1 |
| hypomagnesemia mg/dL<br>Phosphorous – | 18Y-64Y | 2545 | 2.3 - <2.5 | 00 100 | |
| hypophosphatemia mg/dL | 101-041 | 2.5-4.5 | 2.3 - <2.5 | 2.0 - < 2.2 | <2.0 |
| hypophosphatemia mg/dc | 65Y-133Y | mg/dL<br>2.1-4.3 | 1.9 - <2.1 | 1.6 – < 1.8 | <1.6 |
| | 051-1551 | mg/dL | 1.9 - \2.1 | 1.0 - < 1.0 | <1.0 |
| CPK – U/L (male) | <196 | Hig/aL | 196 – 1000 | 1001-1500 | >1500 |
| 0. 11 0.2 (maio) | 1.00 | | 100 1000 | 1001-1000 | 7 1000 |
| CPK - U/L (female) | <143 | | 143 – 1000 | 1001-1500 | >1500 |
| Albumin – | 3.6-5.1 g/dL | | 3.0 - 3.5 | 2.7 - 2.9 | <2.7 |
| Hypoalbuminemia g/dL | | | | | |
| Total Protein – | 18Y-19Y | 6.3-8.2 g/dL | 6.1 – 6.3 | 5.7 - 6.0 | <5.7 |
| Hypoproteinemia g/dL | 20Y-133Y | 6.1-8.1 g/dL | 5.9 – 6.1 | 5.5 5.8 | <5.5 |
| Alkaline phosphatase – U/L | 18Y-19Y | 48-230 U/L | 230 – 340 | 341 – 460 | >460 |
| (Male) | 20Y-133Y | 40-115 U/L | 115 – 225 | 226 - 345 | >345 |
| Alkaline phosphatase – U/L | 18Y-19Y | 47-176 U/L | 176 – 286 | 287 – 406 | >406 |
| (Female) | 20Y-49Y | 33-115 U/L | 115 – 225 | 226 – 345 | >345 |
| | 50Y-133Y | 33-130 U/L | 130 – 240 | 241 – 360 | >360 |
| AST (Male) U/L | 18Y-19Y | 12-32 U/L | 32 – 93 | 94 – 163 | >163 |
| Not (Male) or | 20Y-49Y | 10-40 U/L | 40 – 101 | 102 – 171 | >171 |
| | 50Y-133Y | 10-35 U/L | 35 – 96 | 97 – 166 | >166 |
| AST (Female) U/L | 18Y-19Y | 12-32 U/L | 32 – 93 | 94 – 163 | >163 |
| 7.01 (1.011.01.0) 0.12 | 20Y-44Y | 10-30 U/L | 30 – 91 | 92 – 161 | >161 |
| | 45Y-133Y | 10-35 U/L | 35 – 96 | 97 – 166 | >166 |
| ALT (Male) U/L | 18Y-19Y | 8-46 U/L | 46 – 101 | 102 – 171 | >171 |
| (112.0) | 20Y-133Y | 9-46 U/L | 46 - 101 | 102 – 171 | >171 |
| ALT (Female) U/L | 18Y-19Y | 5-32 U/L | 32 - 87 | 88 – 157 | >157 |
| , | 20Y-133Y | 6-29 U/L | 29 – 84 | 85 – 154 | >154 |
| Bilirubin (serum total) | 18Y-19Y | 0.2-1.1 | 1.2 - 1.9 | 2.0 - 2.4 | >2.4 |
| mg/dL | ĺ | mg/dL | | | |
| | 20Y-133Y | 0.2-1.2 | 1.3 – 2.0 | 2.1 – 2.5 | >2.5 |
| | | mg/dL | | | |
| Bilirubin – when ALT ≥105 | | | 1.3 – 1.5 | 1.6 – 2.0 | >2.0 |
| (Hy's law) | 24 404 11 | | 400 477 | 470 070 | > 070 |
| Amylase- U/L | 21 – 101 U/I | <u> </u> | 102 – 177 | 178 – 278 | >278 |
| Lipase- U/L | 7 – 60 U/L | | 60 – 165 | 166 – 250 | >250 |
| Hemoglobin (Male) - g/dL | 18Y | 12.0-16.9 | 11.5 – 12.0 | 10.5 – 11.9 | <10.5 |
| | | g/dL | | | |
| | 19Y-133Y | 13.2-17.1 | 12.7 – 13.2 | 12.2 – 12.7 | <12.2 |
| Llow-riskin (F | 402/ | g/dL | 44.0 44.5 | 0.5 40.0 | 40.5 |
| Hemoglobin (Female) - | 18Y | 11.5-15.3 | 11.0 11.5 | 9.5 10.9 | <9.5 |
| g/dL | 107 1227 | g/dL | 44.0 44.7 | 0.0 14.0 | -0.0 |
| | 19Y-133Y | 11.7-15.5 | 11.2 – 11.7 | 9.8 – 11.2 | <9.8 |
| WBC Increase - cell/mm3 | 18Y | g/dL<br>4,500- | 13,001 – | 17,001 – | >22,000 |
| VVDC IIICIEASE - CEII/IIIIIIS | 101 | 4,500-<br>13,000/uL | 17,000 | 22,000 | ~ZZ,000 |
| | 19Y-133Y | 3,800- | 10,801 – | 14,801 | >19,800 |
| | 131-1331 | 10,800/uL | 14,800 | 19,800 | - 13,000 |
| WBC Decrease - cell/mm3 | 18Y | 4,500- | 3,500 - | 2,500 - | <2,500 |
| 1120 00000000 00000000 | | 13,000/uL | 4,500 | 3,499 | |
| | 19Y-133Y | 3,800- | 2,800 – | 1,800 | <1,800 |
| | | 10,800/uL | 3,800 | 2,799 | , |
| | | | | . , | |

EDSREP 009 T 01 G 

| Lymphocytes Decrease - cell/mm3 | 18Y | 1200-5200<br>cells/uL | 950 – 1,200 | 700 – 949 | <700 |
|---|---|---|---|---|---|
| | 19Y-133Y | 850-3900<br>cells/ul. | 600 – 850 | 450 - 599 | <450 |
| Neutrophils Decrease -<br>cell/mm3 | 18Y | 1800-8000 | 1,300 - | 1,049 – | <1,049 |
| Cell/IIIIIS | 19Y-133Y | cells/uL<br>1500-7800<br>cells/uL | 1,799<br>1,000 –<br>1,499 | 1,299<br>750 – 999 | <750 |
| Eosinophils - cell/mm3 | 15-500 cells/uL | | 500 – 750 | 751 – 1600 | >1600 |
| Platelets Decreased - cell/mm3 | 140,000 - 400,000/ uL | | 130,000 –<br>140,000 | 110,000 -<br>129,999 | <110,000 |
| PT – seconds (prothrombin time) | 9.0-11.5 seconds | | > ULN-14.4 | 14.5 – 15.7 | >15.7 |
| PTT – seconds (partial thromboplastin time) | 22-34 sec | | >ULN-34.1 | 34.2-42.0 | >42.0 |
| Fibrinogen increase - mg/dL | 175-425 mg/dL | | >ULN – 425 | 426 – 525 | >525 |
| Fibrinogen decrease - 175-425 mg/dL mg/dL | | /dL | <lln 175<="" td="" –=""><td>160 – 174</td><td>&lt;160</td></lln> | 160 – 174 | <160 |
| Urine * | | | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe (Grade 3) |
| Protein | | | 1+ | 2+ | >2+ |
| Glucose | | | 1+ | 2+ | >2+ |
| Blood (microscopic) - red<br>blood cells per high power<br>field (rbc/hpf) | | | 5-10 | 11-50 | > 50 and/or gross<br>blood |
| | | | les serve as gui | delines and are | e dependent upon |
| * Institutional normal reference ranges should be provided to demonstrate that they are appropriate. | | | | | |
| ** Reference ranges are from Quest Diagnostics. Any age range that is not specified is 18Y – 133Y | | | | | |


# **Document History**

| Version Date | Modified/Reviewed By | Brief Summary of Changes |
|---|---|---|
| 21-Jan-2018 | Jacqueline Cater<br>Stephannie Kollipara<br>Emily Mick | Created from EDSREP 009 T 01 G. |
| 28-Mar-2018 | Jacqueline Cater<br>Emily Mick | Revised according to sponsor comments (using updated protocol and eCRF). |

EDSREP 009 T 01 G 



# A PHASE 1 DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF GALIDESIVIR (BCX4430) ADMINISTERED AS SINGLE DOSES VIA INTRAVENOUS INFUSION IN HEALTHY SUBJECTS

Protocol #: BCX4430-106 / DMID 18-0013 PRA Study Code: 181392

# **Dose Escalation Report**

Single Ascending Dose

Cohort 1: 5 mg/kg

Report Date: 07Jan2019

For BioCryst:

Bill Sheridan, MB, BS, Medical Monitor / Chief Medical Officer

Amanda Mathis, PhD, Clinical Pharmacologist

DMID:

Venus S. Shahamatdar, MD, Medical Monitor

Kay M. Tomashek, MD, MPH, DTM, Medical Officer

Carol Ostrye, RN, MPH, Clinical Project Manager

For PRA:

Daniel Dickerson, MD, PhD, Principal Investigator

Jamie Easum, APRN-BC, Co-Lead Sub-Investigator

Lesa Davis, PA-C, Co-Lead Sub-Investigator

Traci Goodwin, Clinical Study Manager

Tim Theisen, Project Manager

Safety Assessment Following Dose Administration of BCX4430 or Placebo to Healthy Volunteers
Dose Escalation Report BioCryst BCX4430-106 Version Date: 07Jan2019

## 1.0 Subject Demographics, Dosing Date and Administration Times (All subjects dosed under fed conditions).

| Subject<br># | Screening<br># | MF | Age | Doeing<br>Date | Dosling<br>Time | Discharge from<br>Clinical Site<br>(Date) |
|---|---|---|---|---|---|---|
| m.r.oogn | Ø11-0065 | 100 | 307 | 11Dec 2018 | -0900 | MGDert2000 |
| 11002 | 01-010 | M | 27 | 11Dec2018 | 0906 | 15Dec2018 |
| 11005 | 01-013 | M | 32 | 13Dec2018 | 0900 | 17Dec2018 |
| 11006 | 01-014 | 3.00 | 45 | 13Dec2018 | 0905 | 17Dec2016 |
| 11004 | Q1-012 | F | 42 | 1 SDecaOls | 0190 | 1/Dep2018 |
| 11000 | 01-006 | E | 24 | 1300000018 | C918 | 170000018 |
| 11008 | 01-023 | - F | 52 | 13Dec2018 | 0925 | 17Dec2018 |
| 11007 | 01-029 | F | 32 | 13Dec2018 | 0930 | 17/Dec2018 |

#### 2.0 Adverse Events

| Buildiests<br># | AE<br># | Adverse Event | Diane of<br>Omelet | Time<br>of<br>Oness | Date of<br>Resolution | Time of<br>Resolution | Sevenity | Relationship<br>to IP |
|---|---|---|---|---|---|---|---|---|
| 11007 | 1 | Viral<br>Gashoerteritis | 26Dec2018 | 2100 | 27Dec2018 | 0900 | Mild | Nint related |

#### 2.1 Adverse Event Comments (summarize findings from above table):

| #deject # | AE # | Advante Event | Community |
|---|---|---|---|
| 11007 | 1 | Viral Gastroenteritie | Subject reports on set of nautoes, verniting and diamnos with know exposure to family with viral gastroenteritis over the preceding 26-88 hours. Resolved within 48 hours. |

#### 3.0 Safety Lab Data: (Summary of significant or notable lab results)

| Subj# | Screen<br># | Mill | Age | Laboratory<br>Collection<br>Date | Lab Test | Result | Range | Toxicity<br>Grading |
|---|---|---|---|---|---|---|---|---|
| 11001 | 01-005 | TAT. | 37 | 11Dec2018 | Total Protein | 6.0 g/dL | 61:81 g/dL | 1 |
| 11002 | 01-010 | M | 27 | 31Dec2018 | PT | 12.1 800 | 9.0-11.5 sec | - 1 |
| 11000 | 01-006 | 1 | 24 | :10ec2018 | CPK | 321 UIL | 29-143-0/4 | 1 |
| 11000 | 01:006 | 18 | 24 | 14Dec2018 | CPK | 22010/4 | 25-142 U/L | 1 |
| 11000 | 01/005 | 15 | 24 | 140012018 | Ollubean | t 400<br>mg/dL | 05-139 ing/80. | 1 |
| 11000 | 01-006 | E | 24 | 1504:2018 | CPK | 165 U/L | 29-145/0/2 | 100 |


Dose Escalation Report BioCryst BCX4430-106 Version Date: 07Jan2019

| | | | | | | | version Date; | u/Janzu |
|---|---|---|---|---|---|---|---|---|
| 11/003 | 01-005 | - | 24 | 16Dec2018 | CPK | 152 U/L | 29-143 U/L | 1 |
| 11003 | Ø1-005 | F | 24 | 16Dec2018 | (CIPIK | 150 U/L | 29-143 U/L | 10 |
| 11003 | 01-005 | E | 24 | 021943019 | CPK | 1290 U/L | 29-143-04 | 2 |
| 11003 | 01.005 | F | 24 | 07/(61/2019 | OPK. | Tahending | | |
| 11034 | 41-012 | E | 45 | sederable | Glunder | 89 mg/40 | CO. B.D. Puppell | 2 |
| 11054 | 01-012 | E | 40 | NO DECEMBER | Gnuces | Ca mgrate | 05-129 ing/dL | 3 |
| 11005 | 01-013 | M | 32 | 13Dec2018 | Phosphale | 1.8<br>mg/dL | 2.5-4.5 mg/dL | 3 |
| 11005 | 01-013 | TUT | 32 | 14Dec2018 | Glucose | 142<br>mg/dL | 65-139 mg/dL | .1 |
| 11005 | 01-013 | 765 | 32 | 15Dec2018 | Olucose | 167<br>mg/dL | 65-139 mg/dl. | 2 |
| 11005 | 01-013 | 160 | 32 | 15Dec2018 | Sodium | 134<br>mmgl/L | 13(5-14(5<br>mmol/L | 1 |
| 11005 | 01-013 | MA | 32 | 16Dec2018 | Olucese | 141<br>mg/dL | 65-139 mg/dL | 1 |
| 11005 | 01-013 | na. | 32 | 17Dec2018 | Siedium | 134<br>mmai/L | 135-148<br>mmol/L | 1. |
| 11006 | 01-014 | TAN | 45 | 13Dec2018 | Phosphate | 2.1<br>mg/dL | 2.5-4.5 mg/dl. | 2 |
| 11006 | 01-014 | M | 45 | 14Dec2018 | Phosphate | 2.4<br>mg/dL | 2.5-4.5 mg/dl. | 1 |
| 11006 | 01-014 | М | 45 | 15Dec2018 | Glucose | 148<br>mg/dL | 65-139 mg/dL | 1 |
| 11006 | 01-014 | M | 45 | 15Dec2018 | Phosphale | 2.4<br>mg/dL | 2.5-4.5 mg/dL | 1 |
| 1007 | 01-029 | F | 32 | 14Dec2018 | Glucose | 62 mg/dL | 65-139 mg/dL | 1 |
| 1007 | 01-029 | P | 32 | 02.lan2019 | Hemoglobin | 11.6 g/dL | 11,7-15.5 g/dL | 1 |
| 1007 | 01-029 | F | 32 | 02.lan2019 | CPK | 189 U/L | 29-143 UIL | 1 |
| 11008 | 01-023 | F | 62 | 02Jan2018 | ALT | 32 U/L | 6-29 UIL | -1 |
| 11008 | 01-023 | * | 62 | 02.Jan2018 | Armylasie | 105 U/L | 21-101/L | 1 |

<sup>\*</sup>N.B. Subject 11004 had elevated CPK at screening and on Day -1.

#### 3.1 Actions Taken/Con Meds Administered Related to Adverse Events:

| Subject AE # | Medication | Dose/Unit | Route Start Date | Stop Date | Prescribed for: |
|---|---|---|---|---|---|

Dose Escalation Report BioCryst BCX4430-106 Version Date: 07Jan2019

4.0 Vital Signs Data (summary of clinically significant abnormal vital signs by subject # and time point taken):

| Subject # | Screening # | M/F | Age | Date | Time | Values | Grade |
|-----------|-------------|-----|-----|------|------|--------|-------|
| | | 1 | | | | | N/A |

<sup>\*</sup>There were no vital signs which met the criteria for halting dosing in Section 11,5,2 of the protocol.

**5.0 12-Lead ECG Data (summarize clinically significant abnormal changes by subject # and time point taken):** There were no clinically significant ECG findings, and no ECG parameters met the criteria for halting dosing stated in Section 11.5.2 of the protocol.

**6.0** Physical Examination Data (summarize clinically significant abnormal changes by subject # and time point performed): There were no clinically significant physical exam findings noted,

7.0 Subject Discontinuations: No subjects were discontinued.

8.0 PK Summary (insert tables, appendices as allowed by sponsor, if available):

Subjects in the table below have been anonymized with an alphabet code. Samples collected through 96 hours post-dose were shipped for analysis, and therefore AUC<sub>0-last</sub> in the table below represents 96 hours. Samples were quantifiable through 96 hours in all subjects. The geometric mean(%CV) C<sub>max</sub>, AUC<sub>0-24</sub> and AUC<sub>0-last</sub> were 5540 ng/mL (8), 10850 ng.h/mL (11), and 14530 ng.h/mL (12), respectively.

No PK parameters met halting rules, and overall, the PK following a 5 mg/kg single dose administered by IV infusion was in line with anticipated exposure based on modeling and simulation.

| Subject<br>Code | T ½ (h) | C <sub>max</sub> *<br>(ng/mL) | AUC <sub>0-24h</sub><br>(ng.h/mL) | AUC <sub>0-last</sub><br>(ng.h/mL) | AUC <sub>0-Inf</sub><br>(ng.h/mL | %AUC<br>extrap | Cl<br>(mL/h/kg) | Vz<br>(mL/kg) |
|---|---|---|---|---|---|---|---|---|
| Α | 96.9 | 5420 | 10000 | 13660 | 19440 | 30 | 257 | 35960 |
| В | 55.9 | 4870 | 11270 | 15190 | 18110 | 16 | 276 | 22270 |
| С | 191.6 | 6140 | 11040 | 14390 | 24760 | 42 | 202 | 55830 |
| D | 75.3 | 5510 | 10460 | 13730 | 17110 | 20 | 292 | 31760 |
| E | 170.6 | 5590 | 12910 | 17830 | 31410 | 43 | 159 | 39180 |
| F | 92.9 | 5820 | 9700 | 12860 | 17320 | 26 | 289 | 38680 |
| Geomean | 103.6 | 5540 | 10850 | 14530 | 20810 | 28 | 240 | 35930 |
| %CV | 50.2 | 8 | 11 | 12 | 27 | 38 | 22 | 30 |

<sup>\*</sup>the timepoint for C<sub>max</sub> was taken at the end of the 1-hour infusion




## 9.0 Investigator opinion about safety of IP based upon clinical tolerance of trial during reported period:

Internal review of all available safety data prior to the dose escalation call shows no concerns with proceeding to the next dose level.

#### 10.0 Summary of Discussion at Dose Escalation Call:

Subject 11004 had a grade 2 elevated CPK at her end of study laboratory evaluation. The subject had no physical symptoms associated with this elevated CPK and on review of her previous labs, she had elevated CPK at screening and on Day -1. She is scheduled to have her CPK redrawn today, 07Jan2019. The safety committee had no concerns regarding this laboratory excursion.

Subjects 1105 and 1106 had grade 2 decreases in phosphate which rapidly corrected. Neither subject had signs or symptoms of hypophosphatemia. The safety committee had no concerns regarding these lab excursions. We will continue monitoring for trends.

Based upon safety measures, tolerance, and pharmacokinetic results, the dose of 5 mg/kg was well tolerated. The Safety Committee discussed data and agreed that data supports moving forward with dose escalation without changes to the protocol.





Current Dose Level: 5 mg/kg Next Dose Level: 10 mg/kg

Protocol changes required prior to next dose level administration (e.g. additional safety monitoring)?

Yes ☐ No ☒

Daniel Dickerson, MD, PhD

Principal Investigator

PRA EDS-Lenexa

Triame Son Palmer MD Mr. For Bill Sherd an

Bill Sheridan, MB, BS

**Medical Monitor** 

BioCryst Chief Medical Officer

1 8000

Date

8 Jan 2019

Date

Amanda Mathis

Director, Clinical Pharmacology

Cimanda Malton

**BioCryst Pharmaceuticals** 

8 Jan 2019 Date



# A PHASE 1 DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF GALIDESIVIR (BCX4430) ADMINISTERED AS SINGLE DOSES VIA INTRAVENOUS INFUSION IN HEALTHY SUBJECTS

Protocol #: **BCX4430-106 / DMID 18-0013**PRA Study Code: **181392** 

### **Dose Escalation Report**

Single Ascending Dose

Cohort 2: 10 mg/kg

Report Date: 01Feb2019

For BioCryst:

Diane Gesty-Palmer MD, PhD, Medical Monitor/Senior Medical Director

Amanda Mathis, PhD, Clinical Pharmacologist

DMID:

Venus S. Shahamatdar, MD, Medical Monitor

Kay M. Tomashek, MD, MPH, DTM, Medical Officer

Carol Ostrye, RN, MPH, Clinical Project Manager

For PRA:

Daniel Dickerson, MD, PhD, Principal Investigator

Jamie Easum, APRN-BC, Co-Lead Sub-Investigator

Lesa Davis, PA-C, Co-Lead Sub-Investigator

Traci Goodwin, Clinical Study Manager

Tim Theisen, Project Manager

Safety Assessment Following Dose Administration of BCX4430 or Placebo to Healthy Volunteers



## 1.0 Subject Demographics, Dosing Date and Administration Times (All subjects dosed under fed conditions).

| Subject<br># | Screening<br># | M/F | Age | Dosing<br>Date | Dosing<br>Time | Discharge from<br>Clinical Site<br>(Date) |
|---|---|---|---|---|---|---|
| 12001 | 01-046 | | 25 | 09Jan2019 | -0900 - | 13Jan2019 |
| 12002 | 01-044 | M | 26 | 09Jan2019 | 0905 | 13Jan2019 |
| 12003 | 01-048 | M | 28 | 11Jan2019 | 0900 | 15Jan2019 |
| 12004 | 01-052 | M | 30 | 11Jan2019 | 0906 | 15Jan2019 |
| 12005 | 01-054 | M | 27 | 11Jan2019 | 0910 | 15,Jan2019 |
| 12006 | 01-055 | M | 45 | 11Jan2019 | 0915 | 15,/an2019 |
| 12007 | 01-057 | F | 40 | 16Jan2019 | 0930 | 20./an2019 |
| 12008 | 01-058 | M | 32 | 22Jan2019 | 0900 | 26.lan2019 |

#### 2.0 Adverse Events

| Subject<br># | AE<br># | Adverse<br>Event | Date of<br>Onset | Time of<br>Onset | Date of<br>Resolution | Time of<br>Resolution | Severity | Relationship to IP |
|---|---|---|---|---|---|---|---|---|

#### 2.1 Adverse Event Comments (summarize findings from above table):

| Subject AE # | Adverse Event | Comments |
|--------------|---------------|----------|



#### 3.0 Safety Lab Data: (Summary of significant or notable lab results)

| Sub # | Screen<br># | 141/<br>F | Age | Laboratory<br>Collection<br>Date | Study | Lab Test | Result | Range | Toxicity<br>Grading |
|---|---|---|---|---|---|---|---|---|---|
| 12001 | 01-046 | F | 25 | 09Jan2019 | 1 | Hermorghobim | 11.0 g/dL | 11.7-15.5 gldL | 2 |
| 12001 | 01-045 | F | 25 | 10Jan2019 | 2 | Hemoglobin | 10.9 g/dL | 11.7-15.5 g/dL | 2 |
| 12001 | 01-046 | F | 25 | 11Jan2019 | 3 | Hemoglobin | 11.1 g/dL | 11.7-15.5 g/dL | 2 |
| 12001 | 01-046 | F | 26 | 11Jan2019 | 3 | RBC (UA) | 3-10 /HPF<br>(on menses) | +/= 2 /HPF | , |
| 12001 | 01-046 | F | 25 | 12Jan2019 | 4 | Hemoglobin | 10.7 g/dL | 11.7-15.5 g/dL | 2 |
| 12001 | 01-045 | * | 25 | 12Jan2019 | 4 | RBC (UA) | 3-10 /HPF<br>(on menses) | < | 1 |
| 12001 | 01-046 | * | 25 | 13Jan2019 | 6 | RBC (UA) | 10-20 /HPF<br>(on menses) | 4/= 2 /HPF | 2 |
| 12001 | 01-046 | F | 25 | 13Jan2019 | 5 | Hemoglobin | 11.3 gldL | 11.7-15.5 g/dL | 1 |
| 12001 | 01-046 | | 25 | 219Jan(2019 | . 21 | PT | 11.6 sec | 9.0-11.5 900 | 1 |
| 12002 | 01-044 | M | 216 | 10Jan2019 | 2 | Glucose (fasting) | 58 mg/dL | 65-99 mg/dL | 2 |
| 12003 | 01-048 | TUT | 28 | 12Jan2019 | 2 | Potassium | 5.5 mmol/L | 3.5-5.3 mmol/L | 2 |
| 12003 | 01-048 | TLET | 218 | 15Jan2019 | 5 | PT | 11.7 sec | 9.0-11.5 sec | 1 |
| 12008 | 01-055 | 1.0 | 4.5 | 11Jan2019 | 1 | Hermoglobile | 12.9 g/dL | 13.2-17.1 g/dL | 1 |
| 12000 | 01-055 | 1.0 | 45 | 11Jan2019 | 1 | Hermoglobin | 13.0 g/dL | 13.2-17.1 gldL | 1 |
| 121006 | 01-055 | 1.0 | 48 | 13Jan2019 | 3 | Hemoglobin | 12.8 g/dL | 13.2/17.1 gldL | 1 |
| 1,2009 | 01-055 | (6.0) | 43 | 15Jan2019 | 8 | Hemoglobin | 13.1 g/dL | 13.2-17.1 g/dl. | 1 |
| 12005 | 01-054 | PLFI. | 27 | 15,Jan2019 | 5 | PT | 11.7 600 | 9.0-11.5 sec | 1 |
| 12005 | 01-054 | RA | 27 | 15Jan2019 | 6 | Amylase | 102 LIIL | 21-101 U/L | 1 |
| 12007 | 01.057 | F. | 40 | reversions. | THE R | Glogose (tasting) | 107 mg/dL | 65-99 mg/dl_ | 24 |
| 12007 | 01-057 | F | 40 | 16UanQ019 | - 16 | Callai, m | A S mg/dL | 8.6 10.2 mg/dL | 1 |
| 1 210/07 | 01-057 | F | 40 | 16Jan2019 | 1 | Albumin | 3.5 g/dL | 3.6-6.1 g/dL | 1 |
| 12007 | 01-057 | SE | 40 | 16Uan2019 | 1 | Hermaglagin | 11.6 g/dL | 11.7-15.5 g/dL | 1 |
| 12007 | 01.057 | E | 40 | 19Jan2019 | E.A | Hemogladin | 11.5 g/dl | 11,7-15,5 g/dL | 1 |
| 12007 | 01:057 | F | 40 | 19Jan2019 | A | Glucese (random) | 142 mg/all | 66-139 mg/dl | 100 |
| 12008 | 01-058 | TUE | 3.2 | 22.lan2019 | 1 | Hermoglobin | 12.9 g/dL | 13.2-17.1 g/dL | 1 |
| 12008 | 01-058 | (LI) | 32 | 23Jan2019 | 2 | Heimoglobin | 13.0 g/dL | 13.2-17.1 g/dL | 1 |
| 12008 | 01-058 | TAE. | 32 | 24Jan2019 | 3 | Hermoglobin | 13.0 g/dL | 13.2-17.1 g/dL | 1 |
| 12008 | 01-05/8 | NAT. | 52 | 25Jan2019 | 4 | Hermoglobin | 13.0 g/dL | 13.2-17.1 g/dL | 1 |



#### 3.1 Actions Taken/Con Meds Administered Related to Adverse Events:



4.0 Vital Signs Data (summary of clinically significant abnormal vital signs by subject # and time point taken):



**5.0 12-Lead ECG Data (summarize clinically significant abnormal changes by subject # and time point taken):** There were no clinically significant ECG findings, and no ECG parameters met the criteria for halting the infusion stated in Section 7.6.3.2 of the protocol.

6.0 Physical Examination Data (summarize clinically significant abnormal changes by subject # and time point performed): There were no clinically significant physical exam findings noted.

7.0 Subject Discontinuations: There were no subject discontinuations throughout this Cohort.

#### 8.0 PK Summary (insert tables, appendices as allowed by sponsor, if available):

Subjects in the table below have been anonymized with an alphabet code. Given the way the cohort dosing was staggered and that samples through only 24 hours post dosing were available for one subject in the cohort, only geometric mean data is presented in order to maintain the blind. If the subject received active, their half-life and clearance parameters are not included in the mean.

Additionally, the  $C_{\text{max}}$  for 3 subjects was greater than 10000 ng/mL (the upper limit of quantitation in the assay) and there was not time to re-assay prior to the dose escalation meeting. Therefore, it is possible that the AUC and  $C_{\text{max}}$  parameters are slightly underestimated. The anticipated geometric mean  $C_{\text{max}}$  for this cohort was approximately 10000-11000 ng/mL, so it is not anticipated that the  $C_{\text{max}}$  concentrations are much greater than 10000 ng/mL, or that the AUC parameters are significantly higher than calculated below.

No PK parameters met halting rules, and overall, the PK following a 10 mg/kg single dose administered by IV infusion was in line with anticipated exposure based on modeling and simulation and the exposure in Cohort 1 (5 mg/kg dose). Furthermore, the simulated exposure for the next two dose levels is not anticipated to exceed the PK stopping criteria in the protocol.

| out y | T ½ (h) | C <sub>max</sub> *<br>(ng/mL) | AUC <sub>0-24h</sub><br>(ng.h/mL) | AUC <sub>0-last</sub><br>(ng.h/mL) | AUC <sub>0-inf</sub><br>(ng.h/mL | %AUC<br>extrap | CI<br>(mL/h/kg) | Vz<br>(mL/kg) |
|---|---|---|---|---|---|---|---|---|
| Geomean | 89.1 | 9240 | 20400 | 30200 | 32400 | 11.1 | 285 | 36600 |
| %CV | 21.6 | 10.6 | 12.8 | 14.1 | 20.9 | 41.5 | 14.2 | 35.4 |

<sup>\* 3</sup> subjects had a Cmax > 10000 ng/mL




The figure below shows the mean galidesivir concentration-time profiles for the first two cohorts of this study.



#### 9.0 Summary of Discussion at Dose Escalation Call:

Based upon safety measures, tolerance, and pharmacokinetic results, the dose of 10 mg/kg was well tolerated. The Safety Committee discussed data and agreed that data supports moving forward with dose escalation and with no change to the protocol.

Current Dose Level: 10 mg/kg
Next Dose Level: 15 mg/kg

Protocol changes required prior to next dose level administration (e.g. additional safety monitoring)?

Yes

No 🖂





Daniel Dickerson, MD, PhD

Principal Investigator

PRA EDS-Lenexa

04 Feb 2019

Diane Som Palma

Diane Gesty-Palmer, MD, PhD

**Medical Monitor** 

BioCryst Sr. Medical Director

01 Feb 2019

Date

Amanda Mathis, PhD

Director, Clinical Pharmacology

**BioCryst Pharmaceuticals** 

01 Feb 2019

Date



# A PHASE 1 DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF GALIDESIVIR (BCX4430) ADMINISTERED AS SINGLE DOSES VIA INTRAVENOUS INFUSION IN HEALTHY SUBJECTS

Protocol #: BCX4430-106 / DMID 18-0013 PRA Study Code: 181392

### **Dose Escalation Report**

Single Ascending Dose

Cohort 3: 15 mg/kg

Report Date: 25Feb2019

For BioCryst: Diane Gesty-Palmer MD, PhD, Medical Monitor/Senior Medical Director

Amanda Mathis, PhD, Clinical Pharmacologist

**DMID:** Venus S. Shahamatdar, MD, Medical Monitor

Kay M. Tomashek, MD, MPH, DTM, Medical Officer

Carol Ostrye, RN, MPH, Clinical Project Manager

For PRA: Daniel Dickerson, MD, PhD, Principal Investigator

Jamie Easum, APRN-BC, Co-Lead Sub-Investigator

Lesa Davis, PA-C, Co-Lead Sub-Investigator

Traci Goodwin, Clinical Study Manager

Tim Theisen, Project Manager

Safety Assessment Following Dose Administration of BCX4430 or Placebo to Healthy Volunteers



## 1.0 Subject Demographics, Dosing Date and Administration Times (All subjects dosed under fed conditions).

| Subject<br># | Screening<br># | M/F | Age | Dosing<br>Date | Dosing<br>Time | Discharge from<br>Clinical Site<br>(Date) |
|---|---|---|---|---|---|---|
| 13001 | 01-064 | М | 32 | 05Feb2019 | 0930 | 09Feb2019 |
| 13002 | 01-071 | F | 28 | 05Feb2019 | 0935 | 09Feb2019 |
| 13003 | 01-078 | М | 27 | 07Feb2019 | 0930 | 11Feb2019 |
| 13004 | 01-080 | М | 54 | 07Feb2019 | 0935 | 11Feb2019 |
| 13005 | 01-088 | М | 54 | 07Feb2019 | 0940 | 11Feb2019 |
| 13006 | 01-082 | F | 34 | 07Feb2019 | 0945 | 11Feb2019 |
| 13007 | 01-089 | F | 49 | 07Feb2019 | 0950 | 11Feb2019 |
| 13008 | 01-090 | F | 37 | 07Feb2019 | 0955 | 11Feb2019 |

#### 2.0 Adverse Events

| Subject<br># | AE<br># | Adverse<br>Event | Date of<br>Onset | Time<br>of<br>Onset | Date of<br>Resolution | Time of<br>Resolution | Severity | Relationship to<br>IP |
|---|---|---|---|---|---|---|---|---|
| 13001 | 1 | Back Pain | 06Feb2019 | 1900 | 08Feb2019 | 0730 | Mild | Not Related |
| 13002 | 1 | Postnasal<br>Drip | 05Feb2019 | 1530 | 11Feb2019 | 0800 | Mild | Not Related |
| 13003 | 1 | Headache | 07Feb2019 | 1700 | 08Feb2019 | 0130 | Mild | Possibly |
| 13005 | -1 | Abdominal<br>Bloating | 10Feb2019 | 0700 | | | Mild | Not Related |
| 13005 | 2 | Nausea | 10Feb2019 | 0700 | 13Feb2019 | 2000 | Mild | Not Related |
| 13005 | 3 | Anorexia | 10Feb2019 | 0700 | | | Mild | Not Related |
| 13007 | 1 | Headache | 07Feb2019 | 1355 | 10Feb2019 | 0545 | Mild | Possibly |
| 13007 | 2 | Vomiting | 08Feb2019 | 0851 | 08Feb2019 | 0852 | Mild | Not Related |
| 13007 | .3 | Syncope | 13Feb2019 | 1330 | 13Feb2019 | 1310 | Mild | Not Related |
| 13007 | 4 | Right Wrist<br>Pain | 13Feb2019 | 1330 | | | Mild | Not Related |
| 13008 | 5 | Urticaria | 20Feb2019 | 1600 | | | Mild | Not Related |
| 13008 | 1 | Headache | 07Feb2019 | 0900 | 10Feb2019 | 1900 | Mild | Not Related |



#### 2.1 Adverse Event Comments (summarize findings from above table):

| Subject | AE<br># | Adverse Event | Comments |
|---|---|---|---|
| 13001 | 1 | Back Pain | Subject complains of aching lumbar back pain secondary to laying in bed. Initially pain rated 6/10 and after adding pillows to lumbar area and heating pad, pain decreased to 3/10. No treatment required. |
| 13002 | 1 | Postnasal Drip | Subject complains of scratchy/itchy/sore throat with accompanying dry cough. No other associated symptoms. Humidifier placed in room and advised increased PO fluids. No treatment required. |
| 13003 | Headache | | Subject complains of aching frontal headache rated 5/10 with no associated symptoms. No medications were required. |
| 13005 | 3005 1 Abdominal Bloating | | Subject complains of abdominal bloating causing pain and discomfort rated 5-7/10. States normal bowel movements but unable to pass gas. Subject states diet here is very different than his usual diet at home where he predominantly eats a low fat diet. Abdominal exam showed positive bowel sounds, tenderness on palpation and tympanic percussion sounds noted in all quadrants. Advised increased ambulation. Continuing to improve as of 20Feb2019. |
| 13005 | 2 | Nausea | Subject states continuous nausea. Smell of food intensifies feelings of nausea. Subject did not consume any food on 10Feb2019 or 11Feb2019. Nausea resolved 13Feb2019. |
| 13005 | 3 | Anorexia | Subject states complete lack of appetite. Subject did not consume any food on 10Feb2019 or 11Feb2019. Appetite improving as of 20Feb2019. |
| 13007 | 1 | Headache | Subject complains of mild, dull, aching frontal headache rated 1/10 on pain scale. Advised ice pack and increased hydration. No medications were required. |
| 13007 | 2 | Vomiting | Subject vomited approximately 30cc of clear liquid. Subject states that she had just finished drinking 48 ounces of water and "it just came back up". No nausea or abdominal pain preceded the vomiting and subject proceeded to eat breakfast immediately after episode. |
| 13007 | 3 | Syncope | Subject states white taking a shower at home she briefly felt lightheaded and then "woke up on the floor". She states she "was only out for a minute". She denies preceding nausea, headache, visual changes or other associated symptoms. She states she felt fine after "waking up". Neuro exam normal at follow up. |
| 13007 | 4 | Right Wrist Pain | Subject fell on right wrist due to syncopal episode in shower. States pain at rest 1/10 and pain with movement 5-6/10. Physical exam showed pain on palpation predominately on dorsal surface, pain on flexion, extension and lateral movement of wrist. Swelling and ecchymosis noted on exam. Subject sent for xrays of wrist. Subject did not complete x-rays due to her personal choice. She reported |
| | | | improvement in swelling and pain with ability to use fully on 20Feb2019. Will monitor. |
| 13007 | 5 | Urticaria | Subject noticed itching around left axilla and shoulder blade region initially, then later noticed "rash" while looking in the mirror. On exam, 7 lesions with wheal/flare response noted (right 4th proximal phalynx, left axilla, 4 X infrascapular region and 1 X inframedial scapula). Lesions are approximately 15-25mm with increase flare to 40mm and wheals approximately 15-20mm after scratching. Subject states ate shrimp for lunch approximately 2.5-3 hours prior to noticing lesions. No oral or respiratory symptoms. Photos taken. |

EDSEXE 013 T 01 C 

Note: The above information serves to document the review of safety information for the referenced study. The information contained in or appended to this report is not considered a source document and has not been subjected to definitive monitoring

Strictly Confidential. © 2004-2014, PRA Health Sciences. All rights reserved.



13008 1 Headache Subject complained of bitemporal headache rated 5/10, at onset, which decreased to 1-2/10 shortly after that. No associated symptoms and no medications were required for treatment.

#### 3.0 Safety Lab Data: (Summary of significant or notable lab results)

| Sub# | Screen<br># | M/<br>F | Age | Laboratory<br>Collection<br>Date | Study<br>Day | Lab Test | Result | Range | Toxicity<br>Grading |
|---|---|---|---|---|---|---|---|---|---|
| 13001 | 01-064 | M | 32 | 07Feb2019 | 3 | Glucose<br>(random) | 148 mg/dL | 65-139 mg/dL | 1 |
| 13001 | 01-064 | M | 32 | 08Feb2019 | 4 | Glucose<br>(random) | 142 mg/dL | 65-139 mg/dL | 1 |
| 13002 | 01-071 | F | 28 | 05Feb2019 | 1 | Glucose | 100 mg/dL | 65-99 mg/dL | 1 |
| 13002 | 01-071 | F | 28 | 07Feb2019 | 3 | Glucose<br>(random) | 144 mg/dL | 65-139 mg/dL | 1 |
| 13003 | 01-078 | M | 27 | 07Feb2019 | 1 | Total Protein | 6.0 g/dL | 6.1-8.1 g/dL | 1 |
| 13003 | 01-078 | M | 27 | 10Feb2019 | 4 | Glucose<br>(random) | 171 mg/dL | 65-139 g/dL | 2 |
| 13004 | 01-080 | M | 54 | 07Feb2019 | 1 | Albumin | 3.5 g/dL | 3.6-5.1 g/dL | 1 |
| 13004 | 01-080 | M | 54 | 08Feb2019 | 2 | Glucose<br>(random) | 155 mg/dL | 65-139 mg/dL | 1 |
| 13004 | 01-080 | M | 54 | 09Feb2019 | 3 | Glucose<br>(random) | 167 mg/dL | 65-139 mg/dL | 2 |
| 13004 | 01-080 | M | 54 | 10Feb2019 | 4 | Glucose<br>(random) | 144 mg/dL | 65-139 mg/dL | 1 |
| 13004 | 01-080 | M | 54 | 11Feb2019 | 5 | ALT | 47 U/L | 9-46 U/L | 1 |
| 13005 | 01-088 | M | 54 | 07Feb2019 | 1 | Total Protein | 6.0 g/dL | 6.1-8.1 g/dL | 1 |
| 13005 | 01-088 | M | 54 | 08Feb2019 | 2 | Total Protein | 5.8 g/dL | 6.1-8.1 g/dL | 2 |
| 13005 | 01-088 | M | 54 | 08Feb2019 | 2 | Hemoglobin | 12.3 g/dL | 13.2-17.1 g/dL | 2 |
| 13005 | 01-088 | M | 54 | 09Feb2019 | 3 | Glucose<br>(random) | 160 mg/dL | 65-139 mg/dL | 2 |
| 13005 | 01-088 | M | 54 | 09Feb2019 | 3 | Total Protein | 5.6 g/dL | 6,1-8,1 g/dL | 2 |
| 13005 | 01-088 | M | 54 | 09Feb2019 | 3 | Hemoglobin | 12.5 g/dL | 13.2-17.1 g/dL | 2 |
| 13005 | 01-088 | M | 54 | 10Feb2019 | 4 | Glucose<br>(random) | 147 mg/dL | 65-139 mg/dL | 1 |
| 13005 | 01-088 | M | 54 | 10Feb2019 | 4 | Sodium | 134 mmol/L | 134-146<br>mmol/L | 1 |
| 13005 | 01-088 | M | 54 | 10Feb2019 | 4 | Total Protein | 5.5 g/dL | 6.1-8.1 g/dL | 2 |
| 13005 | 01-088 | M | 54 | 10Feb2019 | 4 | Hemoglobin | 12.3 g/dL | 13.2-17.1 g/dL | 2 |
| 13005 | 01-088 | M | 54 | 11Feb2019 | 5 | Glucose | 108 mg/dL | 65-99 mg/dL | 2 |
| 13005 | 01-088 | M | 54 | 11Feb2019 | 5 | Total Protein | 5.8 g/dL | 6.1-8.1 g/dL | 2 |

EDSEXE 013 T 01 C 

Note: The above information serves to document the review of safety information for the referenced study. The information contained in or appended to this report is not considered a source document and has not been subjected to definitive monitoring



| 13005 | 01-088 | М | 54 | 11Feb2019 | 5 | Hemoglobin | 12.6 g/dL | 13.2-17.1 g/dL | 2 |
|---|---|---|---|---|---|---|---|---|---|
| 13005 | 01-088 | M | 54 | 11Feb2019 | 5 | WBC | 10.9<br>thousand/uL | 3.8-10.8<br>thousand/uL | 1 |
| 13005 | 01-088 | М | 54 | 13Feb2019 | Unsch | Hemoglobin | 12.4 g/dL | 13.2-17.1 g/dL | 2 |
| 13005 | 01-088 | M | 54 | 21Feb2019 | Unsch | Hemoglobin | 11.6 g/dL | 13.2-17.1 g/dL | 3 |
| 13005 | 01-088 | M | 54 | 21Feb2019 | Unsch | ALT | 72 U/L | 9-46 U/L | 1 |
| 13006 | 01-082 | F | 34 | 07Feb2019 | 1 | Glucose | 114 mg/dL | 65-99 mg/dL | 3 |
| 13006 | 01-082 | F | 34 | 08Feb2019 | 2 | Glucose<br>(random) | 155 mg/dL | 65-139 mg/dL | 1 |
| 13006 | 01-082 | F | 34 | 10Feb2019 | 4 | Glucose<br>(random) | 141 mg/dL | 65-139 mg/dL | 1 |
| 13007 | 01-089 | F | 49 | 07Feb2019 | 1 | Calcium | 8.5 mg/dL | 8.6-10.2 mg/dL | 1 |
| 13007 | 01-089 | F | 49 | 07Feb2019 | 1 | Total Protein | 5.9 g/dL | 6.1-8.1 g/dL | 1 |
| 13007 | 01-089 | F | 49 | 07Feb2019 | 1 | Albumin | 3.5 g/dL | 3.6-5.1 g/dL | 1 |
| 13007 | 01-089 | F | 49 | 07Feb2019 | 1 | Hemoglobin | 11.2 g/dL | 11.7-15.5 g/dL | 1 |
| 13007 | 01-089 | F | 49 | 08Feb2019 | 2 | Total Protein | 5.8 g/dL | 6.1-8.1 g/dL | 2 |
| 13007 | 01-089 | F | 49 | 08Feb2019 | 2 | Hemoglobin | 11.2 g/dL | 11.7-15.5 g/dL | 1 |
| 13007 | 01-089 | F | 49 | 09Feb2019 | 3 | Hemoglobin | 11.5 g/dL | 11.7-15.5 g/dL | 1 |
| 13007 | 01-089 | F | 49 | 10Feb2019 | 4 | Hemoglobin | 11.3 g/dL | 11.7-15.5 g/dL | 1 |
| 13008 | 01-090 | F | 37 | 07Feb2019 | 1 | Calcium | 8.5 mg/dL | 8.6-10.2 mg/dL | 1 |
| 13008 | 01-090 | F | 37 | 07Feb2019 | 1 | Total Protein | 6.0 g/dL | 6.1-8.1 g/dL | 1 |
| 13008 | 01-090 | F | 37 | 08Feb2019 | 2 | RBC (UA) | 10-20 / HPF<br>(on menses) | = 2 /HPF</td <td>2</td> | 2 |

#### 3.1 Actions Taken/Con Meds Administered Related to Adverse Events:

| Subject AE<br>## | Medication | Dose/Unit | Route | Start<br>Date | Stop Date | Prescribed for: |
|---|---|---|---|---|---|---|
| | | | 1,30 | | | |

<sup>\*</sup>There were no actions /con meds administered related to adverse events.

## 4.0 Vital Signs Data (summary of clinically significant abnormal vital signs by subject # and time point taken):

| Subject # | Screening # | M/F | Age | Date | Time | Values | Grade |
|-----------|-------------|-----|-----|------|------|----------|-------|
| | | | . 4 | | | desir de | |

<sup>\*</sup>There were no vital signs which met the criteria for halting dosing in Section 11.5.2 of the protocol.

EDSEXE 013 T 01 C 



**5.0 12-Lead ECG Data (summarize clinically significant abnormal changes by subject # and time point taken):** There were no clinically significant ECG findings, and no ECG parameters met the criteria for halting the infusion stated in Section 7.6.3.2 of the protocol.

6.0 Physical Examination Data (summarize clinically significant abnormal changes by subject # and time point performed): There were no clinically significant physical exam findings noted.

7.0 Subject Discontinuations: There were no subject discontinuations throughout this Cohort.

#### 8.0 PK Summary (insert tables, appendices as allowed by sponsor, if available):

Subjects in the table below have been anonymized with an alphabet code. Samples were quantifiable through 96 hours in all subjects. The geometric mean (%CV) C<sub>max</sub>, AUC<sub>0-24</sub>, and AUC<sub>0-last</sub> were 17700 (16%) ng/mL, 33900 (17%) ng.h/mL, and 44300 (19%) ng.h/mL. No PK parameters met halting rules outlined in the protocol.

| | T ½ (h) | C <sub>max</sub> (ng/mL) | AUC <sub>0-24h</sub><br>(ng.h/mL) | CI (mL/h/kg) | Vz (mL/kg) |
|---|---|---|---|---|---|
| M | 126 | 16500 | 37700 | 220 | 39900 |
| N | 81.2 | 17400 | 32900 | 283 | 33100 |
| 0 | 78 | 21200 | 39600 | 215 | 24200 |
| Р | 76.9 | 18800 | 29900 | 298 | 33000 |
| Q | 74 | 13200 | 25700 | 358 | 38200 |
| R | 64.1 | 20600 | 40200 | 237 | 21900 |
| Geomean | 81.4 | 17700 | 33900 | 264 | 31000 |
| %CV | 26 | 16 | 17 | 21 | 23 |

Geometric mean summary data from all three cohorts are summarized below. Data from Cohort 1 and 2 have been updated to include all quantifiable PK samples, through the follow up period. Exposure has increased roughly proportional to the increase in dose. Therefore, it can be anticipated that for cohort 4, a 20 mg/kg dose of galidesivir administered by IV infusion would result in a C<sub>max</sub> of approximately 24000 ng/mL and an AUC<sub>0-24</sub> of approximately 45000 ng.h/mL, below the stopping criteria (median AUC<sub>0-24</sub> of 52500 ng.h/mL).

| Dose | T ½ (h) | C <sub>max</sub><br>(ng/mL) | AUC <sub>0-24h</sub><br>(ng.h/mL) | AUC <sub>0-last</sub> ·<br>(ng.h/mL) | CI<br>(mL/h/kg) | Vz<br>(mL/kg) |
|---|---|---|---|---|---|---|
| 5 | 110 (40) | 5540 (8) | 10800 (11) | 17100 (24) | 237 (20) | 37700 (13) |
| 10 | 102 (20) | 10300 (21) | 20800 (14) | 32300 (16) | 270 (16) | 39800 (29) |
| 15 | 81.4 (26) | 17700 (16) | 33900 (17) | 44300 (19) | 264 (21) | 31000 (23) |

<sup>\*</sup>Note for cohort 1 and 2, PK has been quantitated through 21 days of sampling. AUC<sub>0-last</sub> represents a longer period than Cohort 3.

EDSEXE 013 T 01 C 



The figure below shows the mean galidesivir concentration-time profiles for the first two cohorts of this study.



#### 9.0 Summary of Discussion at Dose Escalation Call:

Adverse events for subjects 13005 and 13007 were extensively reviewed. Based upon safety measures, tolerance, and pharmacokinetic results, the dose of 15 mg/kg was well tolerated. The Safety Committee discussed data and agreed that data supports moving forward with dose escalation and with no change to the protocol.

Current Dose Level: 15 mg/kg
Next Dose Level: 20 mg/kg

Protocol changes required prior to next dose level administration (e.g. additional safety monitoring)?

Yes ☐ No ☒



Daniel Dickerson, MD, PhD

Principal Investigator

PRA EDS-Lenexa

277eb 2019 Date

Diane En Palme

Diane Gesty-Palmer, MD, PhD

**Medical Monitor** 

BioCryst Sr. Medical Director

Amanda Mathis, PhD

Director, Clinical Pharmacology

**BioCryst Pharmaceuticals** 

2/W/W19



# A PHASE 1 DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF GALIDESIVIR (BCX4430) ADMINISTERED AS SINGLE DOSES VIA INTRAVENOUS INFUSION IN HEALTHY SUBJECTS

Protocol #: **BCX4430-106 / DMID 18-0013**PRA Study Code: **181392** 

### Dose Escalation Report

Single Ascending Dose

Cohort 4: 20 mg/kg

Report Date: 26Mar2019

For BioCryst:

Diane Gesty-Palmer MD, PhD, Medical Monitor/Senior Medical Director

Amanda Mathis, PhD, Clinical Pharmacologist

DMID:

Venus S. Shahamatdar, MD, Medical Monitor

Kay M. Tomashek, MD, MPH, DTM, Medical Officer

Carol Ostrye, RN, MPH, Clinical Project Manager

For PRA:

Daniel Dickerson, MD, PhD, Principal Investigator

Jamie Easum, APRN-BC, Co-Lead Sub-Investigator

Lesa Davis, PA-C, Co-Lead Sub-Investigator

Traci Goodwin, Clinical Study Manager

Tim Theisen, Project Manager

Safety Assessment Following Dose Administration of BCX4430 or Placebo to Healthy Volunteers



## 1.0 Subject Demographics, Dosing Date and Administration Times (All subjects dosed under fed conditions).

| Subject<br># | Screening<br># | M/F | Age | Dosing<br>Date | Dosing<br>Time | Discharge from Clinical<br>Site (Date) |
|---|---|---|---|---|---|---|
| 14001 | 01-126 | М | 39 | 06Mar2019 | 0900 | 10Mar2019 |
| 14002 | 01-124 | M | 45 | 06Mar2019 | 0905 | 10Mar2019 |
| 14003 | 01-151 | F | 25 | 08Mar2019 | 0900 | 12Mar2019 |
| 14006 | 01-134 | .F | 28 | 08Mar2019 | 0905 | 12Mar2019 |
| 14005 | 01-161 | F | 23 | 08Mar2019 | 0910 | 12Mar2019 |
| 14004 | 01-130 | М | 42 | 08Mar2019 | 0915 | 12Mar2019 |
| 14007 | 01-138 | М | 21 | 08Mar2019 | 0920 | 12Mar2019 |
| 14008 | 01-157 | M | 38 | 08Mar2019 | 0925 | 12Mar2019 |

#### 2.0 Adverse Events

| | Subject<br># | AE<br># | Adverse<br>Event | Date of<br>Onset | Time<br>of<br>Onset | Date of<br>Resolution | Time of<br>Resolution | Severity | Relationship to<br>IP |
|---|---|---|---|---|---|---|---|---|---|
| I | 14001 | 1 | Headache | 06Mar2019 | 1200 | 07Mar2019 | 1500 | Mild | Possibly |

#### 2.1 Adverse Event Comments (summarize findings from above table):

| Subject<br># | AE<br># | Adverse Event | Comments |
|---|---|---|---|
| 14001 | 1 | Headache | Subject states intermittent sharp and throbbing pain in frontal and temporal regions. Rates pain 8/10 at its worst. Subject believes it is due to caffeine withdrawal. Advised increased hydration and rest. Pain resolved without medication. |

#### 3.0 Safety Lab Data: (Summary of significant or notable lab results)

| Sub # | Screen<br># | M/<br>F | Age | Laboratory<br>Collection<br>Date | Study<br>Day | Lab Test | Result | Range | Toxicity<br>Grading |
|---|---|---|---|---|---|---|---|---|---|
| 14001 | 01-126 | M | 39 | 06Mar2019 | 1 | Total Protein | 5.4 g/dL | 6.1-8.1 g/dL | 3 |
| 14001 | 01-126 | M | 39 | 06Mar2019 | 1 | Albumin | 3.4 g/dL | 3.6-5.1 g/dL | 1 |
| 14001 | 01-126 | M | 39 | 06Mar2019 | 1 | Hemoglobin | 12.6 g/dL | 13.2-17.1 g/dL | 2 |
| 14001 | 01-126 | M | 39 | 07Mar2019 | 2 | Total Protein | 6.0 g/dL | 6.1-8.1 g/dL | 1 |
| 14001 | 01-126 | M | 39 | 07Mar2019 | 2 | Hemoglobin | 13.1 g/dL | 13.2-17.1 g/dL | 1 |

EDSEXE 013 T 01 C 

Note: The above information serves to document the review of safety information for the referenced study. The information contained in or appended to this report is not considered a source document and has not been subjected to definitive monitoring



| | | | | | | | | | ZOIVIGIZOT |
|---|---|---|---|---|---|---|---|---|---|
| 14001 | 01-126 | М | 39 | 08Mar2019 | 3 | Total Protein | 5.9 g/dL | 6.1-8.1 g/dL | 1 |
| 14001 | 01-126 | M | 39 | 08Mar2019 | 3 | Hemoglobin | 12.9 g/dL | 13.2-17.1 g/dL | 1 |
| 14001 | 01-126 | M | 39 | 09Mar2019 | 4 | Total Protein | 5.9 g/dL | 6.1-8.1 g/dL | 1 |
| 14001 | 01-126 | M | 39 | 09Mar2019 | 4 | Hemoglobin | 12.9 g/dL | 13.2-17.1 g/dL | 1 |
| 14001 | 01-126 | M | 39 | 10Mar2019 | 5 | PT | 11.6 sec | 9.0-11.5 sec | 1 |
| 14001 | 01-126 | M | 39 | 10Mar2019 | 5 | Total Protein | 5.9 g/dL | 6.1-8.1 g/dL | 1 |
| 14002 | 01-124 | M | 45 | 06Mar2019 | 1 | Total Protein | 5.9 g/dL | 6.1-8.1 g/dL | 1 |
| 14002 | 01-124 | M | 45 | 07Mar2019 | 2 | Total Protein | 6.0 g/dL | 6.1-8.1 g/dL | 1 |
| 14002 | 01-124 | M | 45 | 10Mar2019 | 5 | PT | 11.8 sec | 9.0-11.5 sec | 1 |
| 14003 | 01-151 | F | 25 | 08Mar2019 | 1 | Calcium | 8.2 mg/dL | 8.6-10.2 mg/dL | 2 |
| 14003 | 01-151 | F | 25 | 09Mar2019 | 2 | Calcium | 8.5 mg/dL | 8.6-10.2 mg/dL | 1 |
| 14003 | 01-151 | F | 25 | 12Mar2019 | 5 | PT | 11.6 sec | 9.0-11.5 sec | 1 |
| 14006 | 01-134 | F | 28 | 08Mar2019 | 1 | Calcium | 8.5 mg/dL | 8.6-10.2 mg/dL | 1 |
| 14005 | 01-161 | F | 23 | 09Mar2019 | 2 | WBC | 3.1<br>Thousand/uL | 3.8-10.8<br>thousand/uL | 1 |
| 14005 | 01-161 | F | 23 | 10Mar2019 | 3 | WBC | 3.1<br>Thousand/uL | 3.8-10.8<br>thousand/uL | 1 |
| 14005 | 01-161 | F | 23 | 10Mar2019 | 3 | ANC | 1389 cells/uL | 1500-7800<br>cells/uL | 1 |
| 14005 | 01-161 | F | 23 | 11Mar2019 | 4 | WBC | 3.0<br>Thousand/uL | 3.8-10.8<br>thousand/uL | 1 |
| 14005 | 01-161 | F | 23 | 11Mar2019 | 4 | ANC | 1434 cells/uL | 1500-7800<br>cells/uL | 1 |
| 14005 | 01-161 | F | 23 | 12Mar2019 | 5 | PT | 11.6 sec | 9.0-11.5 sec | 1 |
| 14004 | 01-130 | M | 42 | 08Mar2019 | 1 | Absolute<br>Neutrophils | 1163 cells/uL | 1500-7800<br>cells/uL | 1 |
| 14004 | 01-130 | M | 42 | 12Mar2019 | 5 | PT | 12.0 sec | 9.0-11.5 sec | 1 |
| 14007 | 01-138 | М | 21 | 10Mar2019 | 3 | Glucose<br>(random) | 141 mg/dL | 65-139 mg/dL | 1 |
| 14007 | 01-138 | М | 21 | 11Mar2019 | 4 | Glucose<br>(random) | 166 mg/dL | 65-139 mg/dL | 2 |
| 14007 | 01-138 | M | 21 | 12Mar2019 | 5 | PT | 12.4 sec | 9.0-11.5 sec | 1 |
| 14008 | 01-157 | М | 39 | 09Mar2019 | 2 | Glucose<br>(random) | 175 mg/dL | 65-139 mg/dL | 2 |
| 14008 | 01-157 | М | 39 | 10Mar2019 | 3 | Glucose<br>(random) | 170 mg/dL | 65-139 mg/dL | 2 |
| 14008 | 01-157 | М | 39 | 11Mar2019 | 4 | Glucose<br>(random) | 149 mg/dL | 65-139 mg/dL | 1 |



#### 3.1 Actions Taken/Con Meds Administered Related to Adverse Events:

| Subject<br># | AE<br># | Medication | Dose/Unit | Route | Start<br>Date | Stop Date | Prescribed for: |
|---|---|---|---|---|---|---|---|
| and the same of th | , | | | | | | |

<sup>\*</sup>There were no actions /con meds administered related to adverse events.

## 4.0 Vital Signs Data (summary of clinically significant abnormal vital signs by subject # and time point taken):

| Subject # | Screening # | M/F | Age | Date | Time | Values | Grade |
|---|---|---|---|---|---|---|---|
| | Antonio Cara de Cara d | 4:5 | | | | | |

<sup>\*</sup>There were no vital signs which met the criteria for halting dosing in Section 11.5.2 of the protocol.

**5.0 12-Lead ECG Data (summarize clinically significant abnormal changes by subject # and time point taken):** There were no clinically significant ECG findings, and no ECG parameters met the criteria for halting the infusion stated in Section 7.6.3.2 of the protocol.

6.0 Physical Examination Data (summarize clinically significant abnormal changes by subject # and time point performed): There were no clinically significant physical exam findings noted.

7.0 Subject Discontinuations: There were no subject discontinuations throughout this Cohort.

#### 8.0 PK Summary (insert tables, appendices as allowed by sponsor, if available):

Subjects in the table below have been anonymized with an alphabet code. PK presented in this report is based on nominal sampling times. Samples were available through 24 hours in all subjects and were quantifiable through 24 hours. The geometric mean (%CV)  $C_{max}$  and  $AUC_{0-24}$  were 20500 (16%) ng/mL and 44600(13%) ng.h/mL. No PK parameters met halting rules outlined in the protocol.

| | T ½ (h) | C <sub>max</sub> (ng/mL) | AUC <sub>0-24</sub><br>(ng.h/mL) | CI (mL/h/kg) | Vz (mL/kg) |
|---|---|---|---|---|---|
| S | NR | 25500 | 44200 | 382 | 12100 |
| Т | NR | 19900 | 39800 | 487 | 2610 |
| U | NR | 17000 | 42800 | 449 | 2650 |
| V | NR | 19900 | 43900 | 415 | 8110 |
| W | NR | 24100 | 51200 | 357 | 8190 |
| X | NR | 17900 | 46500 | 349 | 13400 |
| Geomean | NR | 20500 | 44600 | 404 | 6490 |
| %CV | | 16.4 | 8.6 | 13.4 | 58 |

EDSEXE 013 T 01 C 

Across cohorts, galidesivir exposure increased roughly proportional to the increase in dose, with a 3.7-fold increase in geometric mean  $C_{max}$  and a 4.1-fold increase in AUC<sub>0-24</sub> with a 4-fold increase in dose.

| Dose | T ½ (h) | C <sub>max</sub><br>(ng/mL) | AUC <sub>0-24</sub><br>(ng.h/mL) | AUC <sub>0-last</sub> •<br>(ng.h/mL) | CI<br>(mL/h/kg) | Vz (mL/kg) |
|---|---|---|---|---|---|---|
| 5 | 110 (40) | 5540 (8) | 10800 (11) | 17100 (24) | 237 (20) | 37700 (13) |
| 10 | 102 (20) | 10300 (21) | 20800 (14) | 32300 (16) | 270 (16) | 39800 (29) |
| 15 | 81.4 (26) | 17700 (16) | 33900 (17) | 59600 (21) | 228 (22) | 56400 (12) |
| 20 | NR | 20500 (16) | 44600 (9) | 44600 (9) | 404 (13) | NR |

<sup>\*</sup>Note for cohort 1,2 and 3, PK has been quantitated through 21 days of sampling. AUC<sub>0-last</sub> represents a longer period than Cohort 3.

The figures below shows the mean galidesivir concentration-time profiles for all cohorts of this study. As Cohort 4 only has PK available through 24 hours, the figure on the right shows concentration-time profiles for all cohorts through 24 hours.



#### 9.0 Summary of Discussion at Dose Escalation Call:

Based upon safety measures, tolerance, and pharmacokinetic results, the dose of 20 mg/kg was well tolerated. The Safety Committee discussed data and agreed that data supports safety of 20 mg/kg dose.

The safety committee reviewed previous SAEs and outstanding AEs:

Subject 12007, in Cohort 2, had a pregnancy that resulted in a spontaneous abortion. Hospital records have been obtained but follow-up gynecologic records were never received. The information was reviewed with the safety committee and the final SAE report will be submitted on 27-Mar-2019. The PI deemed that the SAE was unlikely related to study drug due to subject's age and prior history of spontaneous abortion. The Sponsor concurred that the spontaneous abortion was unlikely related to study drug. In addition, this assessment is consistent with the reported preclinical toxicology.

EDSEXE 013 T 01 C 



Subject 13005, in Cohort 3, reported to the PI on 26-Mar-2019 that he was in the hospital and had a "mass on his stomach". Hospital records are not yet available. The subject had four adverse events on study that are potentially related to his stomach mass. On day 1 of the study (08-Feb-2019) the subject developed anemia which was worked up and found to be an iron deficiency anemia with a negative stool hemoccult, normal reticulocyte count, and low serum iron. On day 3 of the study (10-Feb-2019) he reported abdominal bloating, nausea, and anorexia.

The stomach mass was reported as an SAE on 26-Mar-2019 and the PI deemed it to be unrelated to study drug because potential mass related adverse events began within days after dosing. All members of the safety committee, including the medical monitor, concur with this assessment.

Subject 13007, in Cohort 3, developed urticaria which was evaluated by a dermatologist and found to be vascular urticaria on biopsy. Following dermatology workup, the subject noted working and sleeping at a facility that was found to have bedbugs. The follow-up dermatology report lists bedbugs as consistent with the subject's vascular urticaria. This adverse event was deemed by PI to not be related to study drug based on subject history and dermatology report.

Current Dose Level: 20 mg/kg

Next Dose Level: NA

Protocol changes required prior to next dose level administration (e.g. additional safety monitoring)?

Yes ☐ No ☒

The protocol has completed enrollment of all cohorts and therefore there will be no further doses administered.

This report is intended to summarize the exposure of BCX4430 observed in cohort 4.

There were no stopping criteria met in any cohort of the study

There were no trends or dose relatedness to any laboratory abnormalities.

Overall, galidesivir was well tolerated and has an acceptable safety profile, supporting further clinical development.

EDSEXE 013 T 01 C 



Daniel Dickerson, MD, PhD

Principal Investigator

PRA EDS-Lenexa

28 Mar 2019

Drawe Son Palner

Diane Gesty-Palmer, MD, PhD

Medical Monitor

BioCryst Sr. Medical Director

28 March 2019

Amanda Mathis, PhD

Director, Clinical Pharmacology

unanda Mat

**BioCryst Pharmaceuticals** 

28 March 2019

